CLINICAL TRIAL: NCT00724867
Title: A Multi-Center, Continuation Trial of Belimumab (HGS1006, LymphoStat-B™), a Fully Human Monoclonal Anti-BLyS Antibody, in Subjects With Systemic Lupus Erythematosus (SLE) Who Completed the Phase 3 Protocol HGS1006-C1056 in the United States
Brief Title: A Continuation Trial for Subjects With Lupus Who Completed Protocol HGS1006-C1056 in the United States
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112233; HGS1006-C1066 (Other: Human Genome Sciences)
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Belimumab; SLE; Antibodies; Lupus; Autoimmune Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Belimumab 1 mg/kg (Experimental): Belimumab 1 mg/kg IV every 28 days
  Interventions: Biological: Belimumab 1 mg/kg
- Belimumab 10 mg/kg (Experimental): Belimumab 10 mg/kg IV every 28 days
  Interventions: Biological: Belimumab 10 mg/kg

INTERVENTIONS:
Biological: Belimumab 1 mg/kg — Belimumab 1 mg/kg IV over one hour every 28 days
  Other Names: BENLYSTA; HGS1006; LymphoStat-B™
  Arms: Belimumab 1 mg/kg
Biological: Belimumab 10 mg/kg — Belimumab 10 mg/kg IV over one hour every 28 days
  Other Names: LymphoStat-B™; BENLYSTA; HGS1006
  Arms: Belimumab 10 mg/kg

SUMMARY:
This is a continuation study to provide continuing treatment to subjects who completed study HGS1006-C1056 in the United States, to evaluate the long-term safety and efficacy of belimumab(LymphoStat-B™) in subjects with SLE disease.

DETAILED DESCRIPTION:
This is a long-term continuation study to provide continuing treatment to subjects who completed study HGS1006-C1056 in the United States. This study is to evaluate the long-term safety and efficacy of belimumab (LymphoStat-B™) in subjects with SLE disease.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the HGS1006-C1056 protocol in the United States through Week 72 visit.
* Be able to receive 1st dose of belimumab for HGS 1006-c1066 four weeks after last dose in HGS1006-c1056.

Exclusion Criteria:

* Have developed any other medical disease or condition that has made the subject unsuitable for this study in the opinion of their physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2008-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- United States (46):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Munster, Indiana
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Cumberland, Maryland
  - GSK Investigational Site, Hagerstown, Maryland
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Smithtown, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Arlington, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Onalaska, Wisconsin

REFERENCES:
- [Derived] Strand V, Berry P, Lin X, Asukai Y, Punwaney R, Ramachandran S. Long-Term Impact of Belimumab on Health-Related Quality of Life and Fatigue in Patients With Systemic Lupus Erythematosus: Six Years of Treatment. Arthritis Care Res (Hoboken). 2019 Jun;71(6):829-838. doi: 10.1002/acr.23788. Epub 2019 Apr 29. PMID 30320964
- [Derived] Furie RA, Wallace DJ, Aranow C, Fettiplace J, Wilson B, Mistry P, Roth DA, Gordon D. Long-Term Safety and Efficacy of Belimumab in Patients With Systemic Lupus Erythematosus: A Continuation of a Seventy-Six-Week Phase III Parent Study in the United States. Arthritis Rheumatol. 2018 Jun;70(6):868-877. doi: 10.1002/art.40439. Epub 2018 Apr 25. PMID 29409143

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with systemic lupus erythematosus who completed the Phase 3 HGS1006-C1056 were enrolled to receive belimumab
Groups:
- Belimumab 10 mg/kg IV: Participants, who had received belimumab 1milligram per kilogram (mg/kg) or 10 mg/kg or placebo in study HGS1006-C1056 , received intravenous (IV) infusion of belimumab 10 mg/kg body weight over 1 hour every 28 days. The first dose of belimumab was given 4 weeks (2 to 8 weeks) after the last dose in the HGS1006-C1056 study. Treatment continued for five years from the time the last participant enrolled in the study or until there were 100 or fewer participants enrolled. All participants received standard of care (SoC) for systemic lupus erythematosus (SLE) during study participation.
Period: Overall Study
Arm/Group | Belimumab 10 mg/kg IV
Started | 268
Completed | 140
Not Completed | 128
Not completed — Adverse Event | 25
Not completed — Lack of Efficacy | 14
Not completed — Lost to Follow-up | 12
Not completed — Non-compliance with study drug | 6
Not completed — Physician Decision | 17
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 31
Not completed — Sponsor decision to end study | 14
Not completed — Subject incarcerated | 1
Not completed — Developed withdrawal criteria- pregnancy | 4
Not completed — Subject moved out of state | 1
Not completed — Elected to exit due to site closure | 2

BASELINE CHARACTERISTICS:
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.8 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250
  Male | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American/African Heritage | 57
  American Indian or Alaska Native | 8
  Asian: Central Asian Heritage | 0
  Asian: East Asian Heritage | 2
  Asian: Japanese Heritage | 3
  Asian: South Asian Heritage | 1
  Asian: Southeast Asian Heritage | 7
  Native Hawaiian or Other Pacific Islander | 0
  White: Middle East/North African Heritage | 3
  White: White/Caucasian/European Heritage | 183
  Mixed Race | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Type of Adverse Event (AEs) and Serious Adverse Event (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant (par.) temporally associated with the use of a investigational product (IP), whether or not considered related to the IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of an IP. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is an important medical event that jeopardizes the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, or is associated with liver injury and impaired liver function. Only those participants available at the specified time points (represented by n=X, in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: Modified Intent to Treat (MIIT) Population: The MITT Population comprised of all the participants enrolled in the study who received at least one dose of IP.
Measure: Number; unit: Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Participants
  AE, Any time post baseline, n=268 | 267
  AE, Year 0-1, n=268 | 260
  AE, Year 1-2, n=259 | 235
  AE, Year 2-3, n=244 | 206
  AE, Year 3-4, n=219 | 184
  AE, Year 4-5, n=202 | 167
  AE, Year 5-6, n=192 | 145
  AE, Year 6-7, n=130 | 87
  AE, Year 7 plus, n=65 | 31
  SAE, Any time post baseline, n=268 | 112
  SAE, Year 0-1, n=268 | 33
  SAE, Year 1-2, n=259 | 30
  SAE, Year 2-3, n=244 | 25
  SAE, Year 3-4, n=219 | 22
  SAE, Year 4-5, n=202 | 24
  SAE, Year 5-6, n=192 | 16
  SAE, Year 6-7, n=130 | 13
  SAE, Year 7 plus, n=65 | 3

2. Primary Outcome: AE Rates by System Organ Class (SOC) During the Study
Description: AE rates by SOC adjusting for participant-years on study drug anytime post Baseline are summarized, which included the follow up visits. Only treatment-emergent adverse events (AEs) are summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. The event rate of an AE was calculated as the number of events per 100 participant years: Event Rate = 100* Number of Events / Participant Years. Participant years were calculated as sum across all participants ([last visit of interval day - first visit of interval day + 1]/365). Participant years excluded between study gaps if participant had not started extension study on date of last visit of parent study.
Time Frame: Up Week 440
Population: MITT Population
Measure: Number; unit: Adverse events/100 participant-years
Groups:
- Belimumab 10 mg/kg IV: Participants, who had received belimumab 1mg/kg or 10 mg/kg or placebo in study HGS1006-C1056 , received IV infusion of belimumab 10 mg/kg body weight over 1 hour every 28 days. The first dose of belimumab was given 4 weeks (2 to 8 weeks) after the last dose in the HGS1006-C1056 study. Treatment continued for five years from the time the last participant enrolled in the study or until there were 100 or fewer participants enrolled. All participants received SoC for systemic lupus erythematosus (SLE) during study participation.
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Adverse events/100 participant-years
  Infections and infestations | 134.4
  Musculoskeletal and connective tissue disorders | 75.5
  Gastrointestinal disorders | 53.6
  Injury, poisoning and procedural complications | 32.3
  Skin and subcutaneous tissue disorders | 30
  Nervous system disorders | 29.7
  Respiratory, thoracic and mediastinal disorders | 28.5
  General disorders and administration sitecondition | 27.9
  Psychiatric disorders | 12.4
  Metabolism and nutrition disorders | 10.1
  Vascular disorders | 9.1
  Investigations | 9.1
  Eye disorders | 8.2
  Reproductive system and breast disorders | 6.7
  Cardiac disorders | 6.4
  Immune system disorders | 6
  Renal and urinary disorders | 5.3
  Neoplasms benign, malignant and unspecified | 5
  Blood and lymphatic system disorders | 4.4
  Ear and labyrinth disorders | 3.8
  Hepatobiliary disorders | 2.3
  Endocrine disorders | 1.8
  Social circumstances | 0.8
  Congenital, familial and genetic disorders | 0.5
  Pregnancy, puerperium and perinatal conditions | 0.1

3. Primary Outcome: SAE Rates by System Organ Class (SOC) During the Study
Description: SAE rates by SOC adjusting for participants-years on study drug anytime post Baseline are summarized, which included the follow up visits. Only treatment-emergent SAEs are summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. The event rate of an SAE was calculated as the number of events per 100 participant years: Event Rate = 100* Number of Events / participants Years. participants years were calculated as = sum across all participants ([last visit of interval day - first visit of interval day + 1]/365). participants years excluded between study gaps if participant had not started extension study on date of last visit of parent study.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Number; unit: Adverse events/100 participant-years
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Adverse events/100 participant-years
  Infections and infestations | 4
  Gastrointestinal disorders | 2.2
  Musculoskeletal and connective tissue disorders | 2
  General disorders and administration sitecondition | 1.7
  Nervous system disorders | 1.4
  Injury, poisoning and procedural complications | 1.4
  Vascular disorders | 1
  Neoplasms benign, malignant and unspecified | 1
  Respiratory, thoracic and mediastinal disorders | 0.7
  Cardiac disorders | 0.6
  Metabolism and nutrition disorders | 0.6
  Psychiatric disorders | 0.5
  Renal and urinary disorders | 0.5
  Hepatobiliary disorders | 0.4
  Blood and lymphatic system disorders | 0.3
  Reproductive system and breast disorders | 0.3
  Immune system disorders | 0.1
  Investigations | 0.1
  Skin and subcutaneous tissue disorders | 0.1
  Congenital, familial and genetic disorders | 0.1
  Endocrine disorders | 0.1
  Eye disorders | 0.1
  Pregnancy, puerperium and perinatal conditions | 0.1

4. Primary Outcome: Change From Baseline in Activated Partial Thromboplastin Time (APTT) and Prothrombin Time (PT) at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline (BL) (Day 0), Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion). Change from Baseline in APTT and PT is summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post- Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Seconds
  APTT, Year 1, Week 4, n= 82 | 1.3 (4.46)
  APTT, Year 1, Week 12, n= 79 | 1 (4.56)
  APTT, Year 1, Week 24, n= 243 | 0.7 (4.81)
  APTT, Year 1, Week 36, n= 71 | 1.4 (4.83)
  APTT, Year 1, Week 48, n= 246 | 1.7 (5.37)
  APTT, Year 2, Week 24, n= 231 | 2.7 (5.88)
  APTT, Year 2, Week 48, n= 220 | 3.9 (5.39)
  APTT, Year 3, Week 24, n= 206 | 4.5 (4.92)
  APTT, Year 3, Week 48, n= 202 | 4 (5.34)
  APTT, Year 4, Week 24, n= 201 | 4.2 (6.51)
  APTT, Year 4, Week 48, n= 185 | 4.7 (8.19)
  APTT, Year 5, Week 24, n= 174 | 4.7 (7.03)
  APTT, Year 5, Week 48, n= 171 | 3.6 (5.46)
  APTT, Year 6, Week 24, n= 160 | 4.3 (6.37)
  APTT, Year 6, Week 48, n= 126 | 4.8 (7.71)
  APTT, Year 7, Week 24, n= 118 | 4.4 (4.77)
  APTT, Year 7, Week 48, n= 92 | 5 (9.55)
  APTT, Year 8, Week 24, n= 59 | 4.7 (5.02)
  APTT, Year 8, Week 48, n= 28 | 4.7 (5.51)
  APTT, Year 9, Week 24, n= 2 | 8.5 (13.44)
  APTT, Exit, n= 230 | 3.1 (6.72)
  APTT, 8 Week, Follow-Up, n= 104 | 3.3 (8.58)
  PT, Year 1, Week 4, n= 82 | -0.05 (1.463)
  PT, Year 1, Week 12, n= 79 | -0.66 (3.502)
  PT, Year 1, Week 24, n= 244 | -0.04 (3.239)
  PT, Year 1, Week 36, n= 71 | -0.42 (3.943)
  PT, Year 1, Week 48, n= 246 | 0.2 (4.493)
  PT, Year 2, Week 24, n= 233 | 0.52 (5.059)
  PT, Year 2, Week 48, n= 221 | 0.24 (2.693)
  PT, Year 3, Week 24, n= 206 | 0.26 (2.983)
  PT, Year 3, Week 48, n= 202 | 0.34 (3.77)
  PT, Year 4, Week 24, n= 201 | 0.39 (3.047)
  PT, Year 4, Week 48, n= 186 | 1.96 (14.36)
  PT, Year 5, Week 24, n= 174 | 0.6 (3.56)
  PT, Year 5, Week 48, n= 172 | 0.5 (5.488)
  PT, Year 6, Week 24, n= 160 | 0.39 (3.333)
  PT, Year 6, Week 48, n= 126 | 0.55 (3.473)
  PT, Year 7, Week 24, n= 118 | 0.72 (3.23)
  PT, Year 7, Week 48, n= 92 | 0.68 (5.149)
  PT, Year 8, Week 24, n= 58 | 0.5 (2.401)
  PT, Year 8, Week 48, n= 28 | 1.85 (4.759)
  PT, Year 9, Week 24, n= 2 | 1.45 (2.758)
  PT, Exit, n= 229 | 0.57 (3.972)
  PT, 8 Week, Follow-Up, n= 103 | 0.33 (2.202)

5. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Neutrophils Segmented and Platelets at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline (BL) (Day 0), Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to440 weeks and at follow-up (up to 8 weeks post last infusion). Change from Baseline in basophils, eosinophils, lymphocytes, monocytes, neutrophils, neutrophils segmented and platelets is summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post- Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Billion cells per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Billion cells per liter
  Basophils, Year 1, Week 4, n= 257 | 0.001 (0.0157)
  Basophils, Year 1, Week 12, n= 249 | 0.002 (0.0173)
  Basophils, Year 1, Week 24, n= 249 | 0.003 (0.0175)
  Basophils, Year 1, Week 36, n= 240 | 0.003 (0.0172)
  Basophils, Year 1, Week 48, n= 254 | 0.001 (0.016)
  Basophils, Year 2, Week 24, n= 250 | 0.002 (0.0159)
  Basophils, Year 2, Week 48, n= 233 | 0.001 (0.0157)
  Basophils, Year 3, Week 24, n= 219 | 0.004 (0.0156)
  Basophils, Year 3, Week 48, n= 211 | 0.004 (0.0179)
  Basophils, Year 4, Week 24, n= 210 | 0.004 (0.0157)
  Basophils, Year 4, Week 48, n= 194 | 0.002 (0.0159)
  Basophils, Year 5, Week 24, n= 188 | 0.003 (0.0168)
  Basophils, Year 5, Week 48, n= 184 | 0.005 (0.0226)
  Basophils, Year 6, Week 24, n= 176 | 0.003 (0.0149)
  Basophils, Year 6, Week 48, n= 132 | 0.003 (0.0178)
  Basophils, Year 7, Week 24, n= 122 | 0.005 (0.0189)
  Basophils, Year 7, Week 48, n= 96 | 0.009 (0.0188)
  Basophils, Year 8, Week 24, n= 60 | 0.002 (0.0155)
  Basophils, Year 8, Week 48, n= 29 | 0.002 (0.0147)
  Basophils, Year 9, Week 24, n= 2 | 0.02 (0.0141)
  Basophils, Exit, n= 233 | 0.005 (0.0183)
  Basophils, 8 Week, Follow-Up, n= 106 | 0.004 (0.0186)
  Eosinophils, Year 1, Week 4, n= 257 | -0.001 (0.0893)
  Eosinophils, Year 1, Week 12, n= 249 | 0.005 (0.1089)
  Eosinophils, Year 1, Week 24, n= 249 | 0.008 (0.1281)
  Eosinophils, Year 1, Week 36, n= 240 | 0.004 (0.1279)
  Eosinophils, Year 1, Week 48, n= 254 | 0.007 (0.1216)
  Eosinophils, Year 2, Week 24, n= 250 | 0.006 (0.1228)
  Eosinophils, Year 2, Week 48, n= 233 | -0.009 (0.1234)
  Eosinophils, Year 3, Week 24, n= 219 | -0.002 (0.1303)
  Eosinophils, Year 3, Week 48, n= 211 | -0.023 (0.1276)
  Eosinophils, Year 4, Week 24, n= 210 | -0.034 (0.125)
  Eosinophils, Year 4, Week 48, n= 194 | -0.032 (0.1407)
  Eosinophils, Year 5, Week 24, n= 188 | -0.038 (0.1281)
  Eosinophils, Year 5, Week 48, n= 184 | -0.019 (0.1547)
  Eosinophils, Year 6, Week 24, n= 176 | -0.027 (0.1169)
  Eosinophils, Year 6, Week 48, n= 132 | -0.038 (0.1227)
  Eosinophils, Year 7, Week 24, n= 122 | -0.017 (0.1269)
  Eosinophils, Year 7, Week 48, n= 96 | -0.026 (0.1401)
  Eosinophils, Year 8, Week 24, n= 60 | -0.031 (0.1425)
  Eosinophils, Year 8, Week 48, n= 29 | -0.032 (0.1121)
  Eosinophils, Year 9, Week 24, n= 2 | -0.08 (0.0141)
  Eosinophils, Exit, n= 233 | -0.026 (0.1295)
  Eosinophils, 8 Week, Follow-Up, n= 106 | -0.022 (0.1401)
  Leukocytes, Year 1, Week 4, n= 257 | 0.08 (1.642)
  Leukocytes, Year 1, Week 12, n= 249 | 0.18 (1.856)
  Leukocytes, Year 1, Week 24, n= 249 | -0.02 (1.884)
  Leukocytes, Year 1, Week 36, n= 240 | 0.04 (2.092)
  Leukocytes, Year 1, Week 48, n= 254 | -0.01 (1.863)
  Leukocytes, Year 2, Week 24, n= 250 | -0.19 (2.087)
  Leukocytes, Year 2, Week 48, n= 233 | -0.27 (2.19)
  Leukocytes, Year 3, Week 24, n= 219 | -0.33 (1.959)
  Leukocytes, Year 3, Week 48, n= 211 | -0.42 (1.876)
  Leukocytes, Year 4, Week 24, n= 210 | -0.29 (2.205)
  Leukocytes, Year 4, Week 48, n= 194 | -0.35 (2.207)
  Leukocytes, Year 5, Week 24, n= 188 | -0.4 (2.112)
  Leukocytes, Year 5, Week 48, n= 184 | -0.18 (2.389)
  Leukocytes, Year 6, Week 24, n= 176 | -0.4 (2.161)
  Leukocytes, Year 6, Week 48, n= 132 | -0.24 (2.164)
  Leukocytes, Year 7, Week 24, n= 122 | -0.22 (2.149)
  Leukocytes, Year 7, Week 48, n= 96 | 0.05 (2.388)
  Leukocytes, Year 8, Week 24, n= 60 | 0.17 (2.297)
  Leukocytes, Year 8, Week 48, n= 29 | -0.63 (2.549)
  Leukocytes, Year 9, Week 24, n= 2 | -3.7 (1.273)
  Leukocytes, Exit, n= 233 | 0.09 (2.969)
  Leukocytes, 8 Week, Follow-Up, n= 106 | -0.11 (2.613)
  Lymphocytes, Year 1, Week 4, n= 257 | 0.076 (0.4223)
  Lymphocytes, Year 1, Week 12, n= 249 | 0.039 (0.558)
  Lymphocytes, Year 1, Week 24, n= 249 | 0.002 (0.5023)
  Lymphocytes, Year 1, Week 36, n= 240 | 0.059 (0.5002)
  Lymphocytes, Year 1, Week 48, n= 254 | -0.02 (0.5129)
  Lymphocytes, Year 2, Week 24, n= 250 | -0.073 (0.5033)
  Lymphocytes, Year 2, Week 48, n= 233 | -0.036 (0.5299)
  Lymphocytes, Year 3, Week 24, n= 219 | 0.002 (0.5621)
  Lymphocytes, Year 3, Week 48, n= 211 | -0.028 (0.572)
  Lymphocytes, Year 4, Week 24, n= 210 | -0.036 (0.5809)
  Lymphocytes, Year 4, Week 48, n= 194 | -0.067 (0.5678)
  Lymphocytes, Year 5, Week 24, n= 188 | -0.07 (0.5924)
  Lymphocytes, Year 5, Week 48, n= 184 | -0.047 (0.629)
  Lymphocytes, Year 6, Week 24, n= 176 | -0.021 (0.5876)
  Lymphocytes, Year 6, Week 48, n= 132 | -0.008 (0.5564)
  Lymphocytes, Year 7, Week 24, n= 122 | 0.011 (0.6439)
  Lymphocytes, Year 7, Week 48, n= 96 | 0.143 (0.6619)
  Lymphocytes, Year 8, Week 24, n= 60 | 0.126 (0.6291)
  Lymphocytes, Year 8, Week 48, n= 29 | 0.059 (0.8495)
  Lymphocytes, Year 9, Week 24, n= 2 | 0.765 (1.4354)
  Lymphocytes, Exit, n= 233 | -0.025 (0.6129)
  Lymphocytes, 8 Week, Follow-Up, n= 106 | 0.029 (0.6256)
  Monocytes, Year 1, Week 4, n= 257 | 0.028 (0.1673)
  Monocytes, Year 1, Week 12, n= 249 | 0.036 (0.1694)
  Monocytes, Year 1, Week 24, n= 249 | 0.024 (0.1678)
  Monocytes, Year 1, Week 36, n= 240 | 0.054 (0.1806)
  Monocytes, Year 1, Week 48, n= 254 | 0.044 (0.1754)
  Monocytes, Year 2, Week 24, n= 250 | 0.053 (0.1809)
  Monocytes, Year 2, Week 48, n= 233 | 0.052 (0.1805)
  Monocytes, Year 3, Week 24, n= 219 | 0.059 (0.1809)
  Monocytes, Year 3, Week 48, n= 211 | 0.071 (0.1903)
  Monocytes, Year 4, Week 24, n= 210 | 0.065 (0.1875)
  Monocytes, Year 4, Week 48, n= 194 | 0.084 (0.1782)
  Monocytes, Year 5, Week 24, n= 188 | 0.095 (0.1878)
  Monocytes, Year 5, Week 48, n= 184 | 0.086 (0.1983)
  Monocytes, Year 6, Week 24, n= 176 | 0.072 (0.1826)
  Monocytes, Year 6, Week 48, n= 132 | 0.049 (0.1808)
  Monocytes, Year 7, Week 24, n= 122 | 0.098 (0.1996)
  Monocytes, Year 7, Week 48, n= 96 | 0.097 (0.2032)
  Monocytes, Year 8, Week 24, n= 60 | 0.101 (0.1909)
  Monocytes, Year 8, Week 48, n= 29 | 0.024 (0.2074)
  Monocytes, Year 9, Week 24, n= 2 | 0.03 (0.3818)
  Monocytes, Exit, n= 233 | 0.075 (0.1846)
  Monocytes, 8 Week, Follow-Up, n= 106 | 0.093 (0.1958)
  Neutrophils, Year 1, Week 4, n= 257 | -0.027 (1.6734)
  Neutrophils, Year 1, Week 12, n= 249 | 0.1 (1.7293)
  Neutrophils, Year 1, Week 24, n= 249 | -0.059 (1.8685)
  Neutrophils, Year 1, Week 36, n= 240 | -0.086 (2.1086)
  Neutrophils, Year 1, Week 48, n= 254 | -0.037 (1.7955)
  Neutrophils, Year 2, Week 24, n= 250 | -0.176 (2.0209)
  Neutrophils, Year 2, Week 48, n= 233 | -0.283 (2.1226)
  Neutrophils, Year 3, Week 24, n= 219 | -0.397 (1.8521)
  Neutrophils, Year 3, Week 48, n= 211 | -0.443 (1.763)
  Neutrophils, Year 4, Week 24, n= 210 | -0.288 (2.1214)
  Neutrophils, Year 4, Week 48, n= 194 | -0.342 (2.1425)
  Neutrophils, Year 5, Week 24, n= 188 | -0.392 (1.9654)
  Neutrophils, Year 5, Week 48, n= 184 | -0.207 (2.2312)
  Neutrophils, Year 6, Week 24, n= 176 | -0.424 (2.0787)
  Neutrophils, Year 6, Week 48, n= 132 | -0.251 (2.1415)
  Neutrophils, Year 7, Week 24, n= 122 | -0.315 (2.1382)
  Neutrophils, Year 7, Week 48, n= 96 | -0.176 (2.3755)
  Neutrophils, Year 8, Week 24, n= 60 | -0.025 (2.2303)
  Neutrophils, Year 8, Week 48, n= 29 | -0.681 (2.4214)
  Neutrophils, Year 9, Week 24, n= 2 | -4.44 (0.5798)
  Neutrophils, Exit, n= 233 | 0.058 (2.9836)
  Neutrophils, 8 Week, Follow-Up, n= 106 | -0.214 (2.5793)
  Neutrophils segmented, Year 1, Week 4, n= 257 | -0.028 (1.6685)
  Neutrophils segmented, Year 1, Week 12, n= 249 | 0.098 (1.7212)
  Neutrophils segmented, Year 1, Week 24, n= 249 | -0.059 (1.8683)
  Neutrophils segmented, Year 1, Week 36, n= 240 | -0.086 (2.1097)
  Neutrophils segmented, Year 1, Week 48, n= 254 | -0.044 (1.8014)
  Neutrophils segmented, Year 2, Week 24, n= 250 | -0.177 (2.0163)
  Neutrophils segmented, Year 2, Week 48, n= 233 | -0.284 (2.1204)
  Neutrophils segmented, Year 3, Week 24, n= 219 | -0.397 (1.8509)
  Neutrophils segmented, Year 3, Week 48, n= 211 | -0.444 (1.7607)
  Neutrophils segmented, Year 4, Week 24, n= 210 | -0.286 (2.1249)
  Neutrophils segmented, Year 4, Week 48, n= 194 | -0.342 (2.1464)
  Neutrophils segmented, Year 5, Week 24, n= 188 | -0.39 (1.9703)
  Neutrophils segmented, Year 5, Week 48, n= 184 | -0.207 (2.2273)
  Neutrophils segmented, Year 6, Week 24, n= 176 | -0.422 (2.0826)
  Neutrophils segmented, Year 6, Week 48, n= 132 | -0.249 (2.1432)
  Neutrophils segmented, Year 7, Week 24, n= 122 | -0.313 (2.1378)
  Neutrophils segmented, Year 7, Week 48, n= 96 | -0.179 (2.3698)
  Neutrophils segmented, Year 8, Week 24, n= 60 | -0.025 (2.2303)
  Neutrophils segmented, Year 8, Week 48, n= 29 | -0.681 (2.4214)
  Neutrophils segmented, Year 9, Week 24, n= 2 | -4.44 (0.5798)
  Neutrophils segmented, Exit, n= 233 | 0.046 (2.8796)
  Neutrophils segmented, 8 Week, Follow-Up, n= 106 | -0.215 (2.5788)
  Platelets, Year 1, Week 4, n= 254 | 2.9 (35.71)
  Platelets, Year 1, Week 12, n= 248 | -1.1 (42.04)
  Platelets, Year 1, Week 24, n= 247 | -2 (41.13)
  Platelets, Year 1, Week 36, n= 238 | -5.9 (46.11)
  Platelets, Year 1, Week 48, n= 252 | -8.4 (46.36)
  Platelets, Year 2, Week 24, n= 249 | -17.5 (56.18)
  Platelets, Year 2, Week 48, n= 233 | -18.8 (56.8)
  Platelets, Year 3, Week 24, n= 218 | -17 (56.86)
  Platelets, Year 3, Week 48, n= 210 | -22.4 (57.11)
  Platelets, Year 4, Week 24, n= 210 | -14.6 (64.11)
  Platelets, Year 4, Week 48, n= 193 | -17 (60.26)
  Platelets, Year 5, Week 24, n= 188 | -19 (65.99)
  Platelets, Year 5, Week 48, n= 184 | -17.6 (65.69)
  Platelets, Year 6, Week 24, n= 175 | -18.9 (62.88)
  Platelets, Year 6, Week 48, n= 132 | -23.7 (67.73)
  Platelets, Year 7, Week 24, n= 121 | -14 (77.75)
  Platelets, Year 7, Week 48, n= 96 | -24.7 (64.56)
  Platelets, Year 8, Week 24, n= 60 | -30.5 (65.89)
  Platelets, Year 8, Week 48, n= 29 | -40.7 (62.84)
  Platelets, Year 9, Week 24, n= 2 | 37 (83.44)
  Platelets, Exit, n= 233 | -9.4 (59.82)
  Platelets, 8 Week, Follow-Up, n= 106 | -8 (70.29)

6. Primary Outcome: Change From Baseline in Erythrocytes at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline (BL) (Day 0), at Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion). Change from Baseline in erythrocytes is summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post- Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Trillions cells per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Trillions cells per liter
  Erythrocytes, Year 1, Week 4, n= 257 | 0 (0.243)
  Erythrocytes, Year 1, Week 12, n= 249 | 0.01 (0.284)
  Erythrocytes, Year 1, Week 24, n= 250 | 0.04 (0.291)
  Erythrocytes, Year 1, Week 36, n= 240 | 0.03 (0.309)
  Erythrocytes, Year 1, Week 48, n= 254 | 0.06 (0.337)
  Erythrocytes, Year 2, Week 24, n= 249 | 0.06 (0.341)
  Erythrocytes, Year 2, Week 48, n= 233 | 0.04 (0.338)
  Erythrocytes, Year 3, Week 24, n= 219 | 0.06 (0.361)
  Erythrocytes, Year 3, Week 48, n= 211 | 0.04 (0.362)
  Erythrocytes, Year 4, Week 24, n= 210 | 0.03 (0.37)
  Erythrocytes, Year 4, Week 48, n= 194 | 0.07 (0.376)
  Erythrocytes, Year 5, Week 24, n= 189 | 0.08 (0.395)
  Erythrocytes, Year 5, Week 48, n= 184 | 0.1 (0.412)
  Erythrocytes, Year 6, Week 24, n= 176 | 0.13 (0.405)
  Erythrocytes, Year 6, Week 48, n= 132 | 0.19 (0.393)
  Erythrocytes, Year 7, Week 24, n= 122 | 0.2 (0.438)
  Erythrocytes, Year 7, Week 48, n= 96 | 0.19 (0.441)
  Erythrocytes, Year 8, Week 24, n= 60 | 0.25 (0.404)
  Erythrocytes, Year 8, Week 48, n= 29 | 0.39 (0.403)
  Erythrocytes, Year 9, Week 24, n= 2 | 0.1 (0)
  Erythrocytes, Exit, n= 233 | 0.26 (0.398)
  Erythrocytes, 8 Week, Follow-Up, n= 106 | 0.2 (0.415)

7. Primary Outcome: Change From Baseline in Hematocrit at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline (BL) (Day 0), Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion). Change from Baseline in hematocrit is summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post- Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Percentage
  Hematocrit, Year 1, Week 4, n= 257 | 0.16 (2.247)
  Hematocrit, Year 1, Week 12, n= 249 | 0.11 (2.62)
  Hematocrit, Year 1, Week 24, n= 250 | 0.31 (2.683)
  Hematocrit, Year 1, Week 36, n= 240 | 0.2 (2.836)
  Hematocrit, Year 1, Week 48, n= 254 | 0.73 (3.087)
  Hematocrit, Year 2, Week 24, n= 249 | 0.81 (3.321)
  Hematocrit, Year 2, Week 48, n= 233 | 1.09 (3.433)
  Hematocrit, Year 3, Week 24, n= 219 | 1.4 (3.604)
  Hematocrit, Year 3, Week 48, n= 211 | 1.53 (3.545)
  Hematocrit, Year 4, Week 24, n= 210 | 1.39 (3.448)
  Hematocrit, Year 4, Week 48, n= 194 | 1.67 (3.414)
  Hematocrit, Year 5, Week 24, n= 189 | 1.78 (3.596)
  Hematocrit, Year 5, Week 48, n= 184 | 1.98 (3.943)
  Hematocrit, Year 6, Week 24, n= 176 | 2.16 (3.94)
  Hematocrit, Year 6, Week 48, n= 132 | 2.49 (3.561)
  Hematocrit, Year 7, Week 24, n= 122 | 2.34 (4.166)
  Hematocrit, Year 7, Week 48, n= 96 | 1.86 (4.108)
  Hematocrit, Year 8, Week 24, n= 60 | 2.68 (3.807)
  Hematocrit, Year 8, Week 48, n= 29 | 3.49 (3.554)
  Hematocrit, Year 9, Week 24, n= 2 | 0.7 (0.99)
  Hematocrit, Exit, n= 233 | 3.25 (3.613)
  Hematocrit, 8 Week, Follow-Up, n= 106 | 3.04 (3.478)

8. Primary Outcome: Change From Baseline in Hemoglobin at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline (BL) (Day 0), Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion). Change from Baseline in hemoglobin is summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post- Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Grams per liter
  Hemoglobin, Year 1, Week 4, n= 257 | 0 (7.03)
  Hemoglobin, Year 1, Week 12, n= 249 | 0.3 (8.17)
  Hemoglobin, Year 1, Week 24, n= 250 | 0.5 (8.81)
  Hemoglobin, Year 1, Week 36, n= 240 | 0.5 (9.51)
  Hemoglobin, Year 1, Week 48, n= 254 | 2.1 (10.2)
  Hemoglobin, Year 2, Week 24, n= 250 | 2.5 (11.07)
  Hemoglobin, Year 2, Week 48, n= 233 | 2.4 (11.76)
  Hemoglobin, Year 3, Week 24, n= 219 | 3.7 (11.93)
  Hemoglobin, Year 3, Week 48, n= 211 | 3.9 (11.86)
  Hemoglobin, Year 4, Week 24, n= 210 | 2.5 (11.91)
  Hemoglobin, Year 4, Week 48, n= 194 | 3.2 (11.82)
  Hemoglobin, Year 5, Week 24, n= 189 | 3.7 (12.44)
  Hemoglobin, Year 5, Week 48, n= 184 | 3.7 (13.71)
  Hemoglobin, Year 6, Week 24, n= 176 | 3.7 (13.6)
  Hemoglobin, Year 6, Week 48, n= 132 | 4.2 (13.13)
  Hemoglobin, Year 7, Week 24, n= 122 | 3.3 (14.73)
  Hemoglobin, Year 7, Week 48, n= 96 | 2.6 (14.98)
  Hemoglobin, Year 8, Week 24, n= 60 | 5.2 (12.78)
  Hemoglobin, Year 8, Week 48, n= 29 | 8.4 (12.98)
  Hemoglobin, Year 9, Week 24, n= 2 | -3 (2.83)
  Hemoglobin, Exit, n= 233 | 7.2 (12.46)
  Hemoglobin, 8 Week, Follow-Up, n= 106 | 6.5 (11.93)

9. Primary Outcome: Change From Baseline in Albumin and Protein at the Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline (BL) (Day 0), at Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion). Change from Baseline in albumin and protein is summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post- Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Grams per liter
  Albumin, Year 1, Week 4, n= 251 | -0.3 (2.17)
  Albumin, Year 1, Week 12, n= 248 | 0.1 (2.53)
  Albumin, Year 1, Week 24, n= 246 | 0.3 (2.47)
  Albumin, Year 1, Week 36, n= 238 | 0.4 (2.69)
  Albumin, Year 1, Week 48, n= 250 | 1.1 (2.88)
  Albumin, Year 2, Week 24, n= 248 | 1.1 (3.18)
  Albumin, Year 2, Week 48, n= 233 | 1.2 (3.25)
  Albumin, Year 3, Week 24, n= 218 | 1.3 (3.41)
  Albumin, Year 3, Week 48, n= 209 | 1.4 (3.65)
  Albumin, Year 4, Week 24, n= 207 | 1.3 (3.6)
  Albumin, Year 4, Week 48, n= 194 | 1.5 (3.5)
  Albumin, Year 5, Week 24, n= 184 | 1.7 (3.76)
  Albumin, Year 5, Week 48, n= 178 | 2 (3.69)
  Albumin, Year 6, Week 24, n= 175 | 1.8 (4.05)
  Albumin, Year 6, Week 48, n= 134 | 1.8 (4.09)
  Albumin, Year 7, Week 24, n= 123 | 1.4 (4.14)
  Albumin, Year 7, Week 48, n= 97 | 1.6 (4.19)
  Albumin, Year 8, Week 24, n= 60 | 2 (4.4)
  Albumin, Year 8, Week 48, n= 28 | 2.9 (3.92)
  Albumin, Year 9, Week 24, n= 2 | 1 (0)
  Albumin, Exit, n= 235 | 2.2 (3.59)
  Albumin, 8 Week, Follow-Up, n= 107 | 1.8 (3.77)
  Protein, Year 1, Week 4, n= 251 | -1.3 (3.73)
  Protein, Year 1, Week 12, n= 248 | -1.9 (4.41)
  Protein, Year 1, Week 24, n= 246 | -2.1 (4.31)
  Protein, Year 1, Week 36, n= 238 | -2.6 (4.59)
  Protein, Year 1, Week 48, n= 250 | -1.8 (4.91)
  Protein, Year 2, Week 24, n= 248 | -2.2 (4.9)
  Protein, Year 2, Week 48, n= 233 | -2.6 (5.08)
  Protein, Year 3, Week 24, n= 218 | -2.6 (5)
  Protein, Year 3, Week 48, n= 209 | -3 (5.36)
  Protein, Year 4, Week 24, n= 207 | -3.4 (5.3)
  Protein, Year 4, Week 48, n= 194 | -3.6 (5.22)
  Protein, Year 5, Week 24, n= 184 | -3.4 (5.44)
  Protein, Year 5, Week 48, n= 178 | -3.4 (5.16)
  Protein, Year 6, Week 24, n= 175 | -4 (5.55)
  Protein, Year 6, Week 48, n= 134 | -3.5 (5.81)
  Protein, Year 7, Week 24, n= 123 | -4.3 (5.56)
  Protein, Year 7, Week 48, n= 97 | -4.3 (5.87)
  Protein, Year 8, Week 24, n= 60 | -4.1 (5.78)
  Protein, Year 8, Week 48, n= 28 | -3 (5.18)
  Protein, Year 9, Week 24, n= 2 | -1.5 (2.12)
  Protein, Exit, n= 235 | -2.6 (5.53)
  Protein, 8 Week, Follow-Up, n= 107 | -3.1 (6.19)

10. Primary Outcome: Change From Baseline in Blood Urea Nitrogen, Glucose, Calcium, Carbon Dioxide, Chloride, Magnesium, Phosphate, Potassium and Sodium at the Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline (BL) (Day 0), at Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion). Change from Baseline in blood urea nitrogen, glucose, calcium, carbon dioxide, chloride, magnesium, phosphate, potassium and sodium is summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post- Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Millimoles per liter
  Blood urea nitrogen, Year 1, Week 4, n= 251 | 0.026 (1.4283)
  Blood urea nitrogen, Year 1, Week 12, n= 248 | -0.1695 (1.4782)
  Blood urea nitrogen, Year 1, Week 24, n= 246 | -0.1612 (1.9011)
  Blood urea nitrogen, Year 1, Week 36, n= 238 | -0.1732 (1.5648)
  Blood urea nitrogen, Year 1, Week 48, n= 250 | -0.1013 (1.5557)
  Blood urea nitrogen, Year 2, Week 24, n= 248 | -0.1873 (1.6796)
  Blood urea nitrogen, Year 2, Week 48, n= 233 | -0.0134 (1.7024)
  Blood urea nitrogen, Year 3, Week 24, n= 218 | -0.0552 (1.7117)
  Blood urea nitrogen, Year 3, Week 48, n= 209 | -0.0472 (1.6693)
  Blood urea nitrogen, Year 4, Week 24, n= 207 | -0.09 (1.6775)
  Blood urea nitrogen, Year 4, Week 48, n= 194 | -0.1162 (1.721)
  Blood urea nitrogen, Year 5, Week 24, n= 184 | -0.0331 (1.6526)
  Blood urea nitrogen, Year 5, Week 48, n= 178 | 0.0176 (1.7712)
  Blood urea nitrogen, Year 6, Week 24, n= 175 | -0.0029 (1.6054)
  Blood urea nitrogen, Year 6, Week 48, n= 134 | -0.0858 (1.6972)
  Blood urea nitrogen, Year 7, Week 24, n= 123 | 0.0246 (1.6668)
  Blood urea nitrogen, Year 7, Week 48, n= 97 | -0.008 (1.6683)
  Blood urea nitrogen, Year 8, Week 24, n= 60 | -0.1152 (1.5362)
  Blood urea nitrogen, Year 8, Week 48, n= 28 | -0.1603 (1.5417)
  Blood urea nitrogen, Year 9, Week 24, n= 2 | -0.1805 (1.06)
  Blood urea nitrogen, Exit, n= 235 | 0.0501 (1.7369)
  Blood urea nitrogen, 8 Week, Follow-Up, n= 107 | 0.3248 (2.2109)
  Glucose, Year 1, Week 4, n= 251 | 0.1088 (1.1734)
  Glucose, Year 1, Week 12, n= 248 | 0.2006 (1.1712)
  Glucose, Year 1, Week 24, n= 246 | 0.0881 (1.2279)
  Glucose, Year 1, Week 36, n= 238 | 0.2158 (1.2519)
  Glucose, Year 1, Week 48, n= 250 | 0.1482 (1.5029)
  Glucose, Year 2, Week 24, n= 248 | 0.1146 (1.3072)
  Glucose, Year 2, Week 48, n= 233 | 0.323 (1.5426)
  Glucose, Year 3, Week 24, n= 218 | 0.1927 (1.4319)
  Glucose, Year 3, Week 48, n= 209 | 0.1719 (1.4829)
  Glucose, Year 4, Week 24, n= 207 | 0.2737 (1.6169)
  Glucose, Year 4, Week 48, n= 194 | 0.2523 (2.1698)
  Glucose, Year 5, Week 24, n= 184 | 0.2579 (1.4792)
  Glucose, Year 5, Week 48, n= 178 | 0.2964 (1.7205)
  Glucose, Year 6, Week 24, n= 175 | 0.2903 (1.7746)
  Glucose, Year 6, Week 48, n= 134 | 0.3897 (1.7503)
  Glucose, Year 7, Week 24, n= 123 | 0.297 (2.257)
  Glucose, Year 7, Week 48, n= 97 | 0.5098 (1.8839)
  Glucose, Year 8, Week 24, n= 60 | 0.449 (1.9609)
  Glucose, Year 8, Week 48, n= 28 | 0.7571 (2.2408)
  Glucose, Year 9, Week 24, n= 2 | 0.8845 (0.4094)
  Glucose, Exit, n= 235 | 0.2986 (1.3871)
  Glucose, 8 Week, Follow-Up, n= 107 | 0.3354 (1.4114)
  Calcium, Year 1, Week 4, n= 242 | 0.0071 (0.0888)
  Calcium, Year 1, Week 12, n= 247 | -0.0043 (0.0872)
  Calcium, Year 1, Week 24, n= 244 | -0.0023 (0.0889)
  Calcium, Year 1, Week 36, n= 235 | -0.0156 (0.0884)
  Calcium, Year 1, Week 48, n= 250 | 0.0007 (0.0896)
  Calcium, Year 2, Week 24, n= 246 | -0.0017 (0.0946)
  Calcium, Year 2, Week 48, n= 231 | -0.0019 (0.0922)
  Calcium, Year 3, Week 24, n= 214 | -0.0009 (0.09)
  Calcium, Year 3, Week 48, n= 205 | -0.0109 (0.1004)
  Calcium, Year 4, Week 24, n= 204 | -0.0115 (0.095)
  Calcium, Year 4, Week 48, n= 191 | -0.0072 (0.0889)
  Calcium, Year 5, Week 24, n= 184 | -0.0181 (0.0986)
  Calcium, Year 5, Week 48, n= 176 | -0.0011 (0.0912)
  Calcium, Year 6, Week 24, n= 172 | -0.0107 (0.0977)
  Calcium, Year 6, Week 48, n= 134 | 0.0007 (0.0925)
  Calcium, Year 7, Week 24, n= 121 | 0.0014 (0.0873)
  Calcium, Year 7, Week 48, n= 97 | 0.0063 (0.0964)
  Calcium, Year 8, Week 24, n= 60 | -0.0123 (0.0788)
  Calcium, Year 8, Week 48, n= 28 | 0.0021 (0.0935)
  Calcium, Year 9, Week 24, n= 2 | -0.005 (0.0354)
  Calcium, Exit, n= 235 | 0.0151 (0.0923)
  Calcium, 8 Week, Follow-Up, n= 107 | 0.0046 (0.1029)
  Carbon dioxide, Year 1, Week 4, n= 243 | -0.2 (2.72)
  Carbon dioxide, Year 1, Week 12, n= 245 | -0.4 (2.62)
  Carbon dioxide, Year 1, Week 24, n= 244 | -0.2 (2.51)
  Carbon dioxide, Year 1, Week 36, n= 234 | -0.1 (2.67)
  Carbon dioxide, Year 1, Week 48, n= 250 | -0.2 (2.64)
  Carbon dioxide, Year 2, Week 24, n= 246 | 0 (2.58)
  Carbon dioxide, Year 2, Week 48, n= 231 | -0.5 (2.78)
  Carbon dioxide, Year 3, Week 24, n= 215 | -0.5 (2.75)
  Carbon dioxide, Year 3, Week 48, n= 205 | -0.9 (2.82)
  Carbon dioxide, Year 4, Week 24, n= 204 | -0.6 (2.7)
  Carbon dioxide, Year 4, Week 48, n= 191 | -0.6 (2.79)
  Carbon dioxide, Year 5, Week 24, n= 184 | -0.9 (2.68)
  Carbon dioxide, Year 5, Week 48, n= 176 | -0.7 (2.73)
  Carbon dioxide, Year 6, Week 24, n= 172 | -0.8 (2.62)
  Carbon dioxide, Year 6, Week 48, n= 134 | -0.7 (3.23)
  Carbon dioxide, Year 7, Week 24, n= 121 | -0.7 (2.84)
  Carbon dioxide, Year 7, Week 48, n= 97 | -0.3 (3.14)
  Carbon dioxide, Year 8, Week 24, n= 60 | -0.5 (3.17)
  Carbon dioxide, Year 8, Week 48, n= 28 | -0.7 (2.87)
  Carbon dioxide, Year 9, Week 24, n= 2 | -1 (1.41)
  Carbon dioxide, Exit, n= 235 | 0.1 (2.74)
  Carbon dioxide, 8 Week, Follow-Up, n= 107 | 0 (2.55)
  Chloride, Year 1, Week 4, n= 251 | 0.2 (2.8)
  Chloride, Year 1, Week 12, n= 248 | 0.1 (2.53)
  Chloride, Year 1, Week 24, n= 246 | 0.3 (2.31)
  Chloride, Year 1, Week 36, n= 238 | 0.5 (2.43)
  Chloride, Year 1, Week 48, n= 250 | 0 (2.53)
  Chloride, Year 2, Week 24, n= 248 | 0.1 (2.6)
  Chloride, Year 2, Week 48, n= 233 | 0.1 (3.03)
  Chloride, Year 3, Week 24, n= 218 | -0.1 (3.01)
  Chloride, Year 3, Week 48, n= 209 | 0.1 (3.06)
  Chloride, Year 4, Week 24, n= 207 | -0.4 (3.28)
  Chloride, Year 4, Week 48, n= 194 | -0.3 (2.83)
  Chloride, Year 5, Week 24, n= 184 | -0.3 (3.06)
  Chloride, Year 5, Week 48, n= 178 | -0.1 (3.02)
  Chloride, Year 6, Week 24, n= 175 | 0 (3.11)
  Chloride, Year 6, Week 48, n= 134 | 0.3 (2.89)
  Chloride, Year 7, Week 24, n= 123 | 0.4 (3.1)
  Chloride, Year 7, Week 48, n= 97 | 0.5 (3.28)
  Chloride, Year 8, Week 24, n= 60 | 0.5 (3.21)
  Chloride, Year 8, Week 48, n= 28 | 1.1 (2.49)
  Chloride, Year 9, Week 24, n= 2 | 1.5 (2.12)
  Chloride, Exit, n= 235 | -0.5 (2.96)
  Chloride, 8 Week, Follow-Up, n= 107 | 0.1 (2.65)
  Magnesium, Year 1, Week 4, n= 251 | 0.002 (0.0673)
  Magnesium, Year 1, Week 12, n= 248 | -0.005 (0.0625)
  Magnesium, Year 1, Week 24, n= 246 | 0.004 (0.0599)
  Magnesium, Year 1, Week 36, n= 238 | 0.001 (0.066)
  Magnesium, Year 1, Week 48, n= 250 | 0.001 (0.0677)
  Magnesium, Year 2, Week 24, n= 248 | 0.003 (0.0709)
  Magnesium, Year 2, Week 48, n= 233 | 0.003 (0.0699)
  Magnesium, Year 3, Week 24, n= 218 | 0.007 (0.0719)
  Magnesium, Year 3, Week 48, n= 209 | 0.011 (0.0681)
  Magnesium, Year 4, Week 24, n= 207 | 0.009 (0.0682)
  Magnesium, Year 4, Week 48, n= 194 | 0.012 (0.0692)
  Magnesium, Year 5, Week 24, n= 184 | 0.017 (0.062)
  Magnesium, Year 5, Week 48, n= 178 | 0.014 (0.0622)
  Magnesium, Year 6, Week 24, n= 175 | 0.017 (0.067)
  Magnesium, Year 6, Week 48, n= 134 | 0.003 (0.0664)
  Magnesium, Year 7, Week 24, n= 123 | 0.004 (0.0691)
  Magnesium, Year 7, Week 48, n= 97 | 0.001 (0.0681)
  Magnesium, Year 8, Week 24, n= 60 | -0.006 (0.0644)
  Magnesium, Year 8, Week 48, n= 28 | 0.016 (0.0599)
  Magnesium, Year 9, Week 24, n= 2 | 0.02 (0.0283)
  Magnesium, Exit, n= 235 | 0.03 (0.0676)
  Magnesium, 8 Week, Follow-Up, n= 107 | 0.028 (0.0728)
  Phosphate, Year 1, Week 4, n= 251 | 0.0165 (0.1857)
  Phosphate, Year 1, Week 12, n= 248 | -0.0065 (0.1851)
  Phosphate, Year 1, Week 24, n= 246 | 0.0106 (0.2027)
  Phosphate, Year 1, Week 36, n= 238 | -0.0039 (0.1825)
  Phosphate, Year 1, Week 48, n= 250 | 0.0019 (0.1926)
  Phosphate, Year 2, Week 24, n= 248 | -0.0133 (0.2219)
  Phosphate, Year 2, Week 48, n= 233 | 0.0099 (0.1968)
  Phosphate, Year 3, Week 24, n= 218 | 0.0033 (0.2129)
  Phosphate, Year 3, Week 48, n= 209 | 0.0017 (0.221)
  Phosphate, Year 4, Week 24, n= 207 | -0.0022 (0.2145)
  Phosphate, Year 4, Week 48, n= 194 | -0.0102 (0.1765)
  Phosphate, Year 5, Week 24, n= 184 | -0.015 (0.1899)
  Phosphate, Year 5, Week 48, n= 178 | -0.0035 (0.1892)
  Phosphate, Year 6, Week 24, n= 175 | -0.004 (0.2153)
  Phosphate, Year 6, Week 48, n= 134 | -0.0139 (0.2097)
  Phosphate, Year 7, Week 24, n= 123 | 0.0296 (0.1962)
  Phosphate, Year 7, Week 48, n= 97 | 0.031 (0.1875)
  Phosphate, Year 8, Week 24, n= 60 | -0.0223 (0.2186)
  Phosphate, Year 8, Week 48, n= 28 | -0.0054 (0.2093)
  Phosphate, Year 9, Week 24, n= 2 | 0.1467 (0.1893)
  Phosphate, Exit, n= 235 | 0.0161 (0.2151)
  Phosphate, 8 Week, Follow-Up, n= 107 | 0.0438 (0.2131)
  Potassium, Year 1, Week 4, n= 242 | 0.07 (0.407)
  Potassium, Year 1, Week 12, n= 245 | 0.02 (0.412)
  Potassium, Year 1, Week 24, n= 244 | 0.02 (0.409)
  Potassium, Year 1, Week 36, n= 234 | 0.03 (0.427)
  Potassium, Year 1, Week 48, n= 250 | -0.04 (0.413)
  Potassium, Year 2, Week 24, n= 246 | 0.01 (0.42)
  Potassium, Year 2, Week 48, n= 231 | 0.02 (0.426)
  Potassium, Year 3, Week 24, n= 215 | 0.01 (0.418)
  Potassium, Year 3, Week 48, n= 205 | 0.01 (0.466)
  Potassium, Year 4, Week 24, n= 204 | -0.02 (0.409)
  Potassium, Year 4, Week 48, n= 191 | 0.04 (0.417)
  Potassium, Year 5, Week 24, n= 184 | 0 (0.406)
  Potassium, Year 5, Week 48, n= 176 | 0.06 (0.427)
  Potassium, Year 6, Week 24, n= 172 | -0.03 (0.431)
  Potassium, Year 6, Week 48, n= 134 | 0.06 (0.438)
  Potassium, Year 7, Week 24, n= 121 | 0.04 (0.379)
  Potassium, Year 7, Week 48, n= 97 | 0.06 (0.387)
  Potassium, Year 8, Week 24, n= 60 | 0 (0.354)
  Potassium, Year 8, Week 48, n= 28 | 0.1 (0.401)
  Potassium, Year 9, Week 24, n= 2 | 0.05 (0.212)
  Potassium, Exit, n= 235 | 0.11 (0.431)
  Potassium, 8 Week, Follow-Up, n= 107 | 0.07 (0.493)
  Sodium, Year 1, Week 4, n= 251 | 0.4 (2.67)
  Sodium, Year 1, Week 12, n= 248 | 0 (2.67)
  Sodium, Year 1, Week 24, n= 246 | 0.3 (2.02)
  Sodium, Year 1, Week 36, n= 238 | 0.3 (2.46)
  Sodium, Year 1, Week 48, n= 250 | -0.1 (2.06)
  Sodium, Year 2, Week 24, n= 248 | 0 (2.19)
  Sodium, Year 2, Week 48, n= 233 | 0 (2.58)
  Sodium, Year 3, Week 24, n= 218 | -0.1 (2.18)
  Sodium, Year 3, Week 48, n= 209 | 0.4 (2.44)
  Sodium, Year 4, Week 24, n= 207 | 0.2 (2.54)
  Sodium, Year 4, Week 48, n= 194 | 0.1 (2.36)
  Sodium, Year 5, Week 24, n= 184 | 0.1 (2.19)
  Sodium, Year 5, Week 48, n= 178 | 0 (2.37)
  Sodium, Year 6, Week 24, n= 175 | 0.1 (2.33)
  Sodium, Year 6, Week 48, n= 134 | 0.3 (2.72)
  Sodium, Year 7, Week 24, n= 123 | 0.3 (2.97)
  Sodium, Year 7, Week 48, n= 97 | 0.3 (2.49)
  Sodium, Year 8, Week 24, n= 60 | 0.2 (2.32)
  Sodium, Year 8, Week 48, n= 28 | 0.4 (1.95)
  Sodium, Year 9, Week 24, n= 2 | -1 (1.41)
  Sodium, Exit, n= 235 | 0.1 (2.32)
  Sodium, 8 Week, Follow-Up, n= 107 | 0.8 (2.33)

11. Primary Outcome: Change From Baseline in Creatinine, Urate and Bilirubin at the Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline (BL) (Day 0), at Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion). Change from Baseline in urate, creatinine and bilirubin is summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post- Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Micromoles per liter
  Creatinine, Year 1, Week 4, n= 250 | -0.2 (4.69)
  Creatinine, Year 1, Week 12, n= 248 | -0.5 (4.86)
  Creatinine, Year 1, Week 24, n= 246 | -0.6 (5.31)
  Creatinine, Year 1, Week 36, n= 237 | -0.4 (5.07)
  Creatinine, Year 1, Week 48, n= 250 | -0.2 (5.29)
  Creatinine, Year 2, Week 24, n= 248 | -0.2 (5.76)
  Creatinine, Year 2, Week 48, n= 233 | 0.3 (4.78)
  Creatinine, Year 3, Week 24, n= 218 | 0.8 (5.63)
  Creatinine, Year 3, Week 48, n= 209 | 0.9 (5.61)
  Creatinine, Year 4, Week 24, n= 207 | 1.2 (5.86)
  Creatinine, Year 4, Week 48, n= 194 | 0.9 (6.05)
  Creatinine, Year 5, Week 24, n= 184 | 1 (5.52)
  Creatinine, Year 5, Week 48, n= 178 | 1.2 (6.49)
  Creatinine, Year 6, Week 24, n= 175 | 1.2 (5.79)
  Creatinine, Year 6, Week 48, n= 134 | 1 (6.38)
  Creatinine, Year 7, Week 24, n= 123 | 1.1 (5.75)
  Creatinine, Year 7, Week 48, n= 97 | 0.7 (5.42)
  Creatinine, Year 8, Week 24, n= 60 | 0.8 (5.09)
  Creatinine, Year 8, Week 48, n= 28 | 0.4 (5.28)
  Creatinine, Year 9, Week 24, n= 2 | -0.5 (0.71)
  Creatinine, Exit, n= 235 | 1.1 (5.57)
  Creatinine, 8 Week, Follow-Up, n= 107 | 1.3 (5.99)
  Urate, Year 1, Week 4, n= 251 | -1.653 (46.0197)
  Urate, Year 1, Week 12, n= 248 | -5.5803 (52.2256)
  Urate, Year 1, Week 24, n= 246 | -11.6488 (55.2277)
  Urate, Year 1, Week 36, n= 238 | -9.984 (57.2999)
  Urate, Year 1, Week 48, n= 250 | -4.108 (58.0533)
  Urate, Year 2, Week 24, n= 248 | -6.4785 (57.0915)
  Urate, Year 2, Week 48, n= 233 | -4.6501 (60.3008)
  Urate, Year 3, Week 24, n= 218 | 1.6919 (63.7367)
  Urate, Year 3, Week 48, n= 209 | -4.5543 (66.183)
  Urate, Year 4, Week 24, n= 207 | -4.8112 (60.2771)
  Urate, Year 4, Week 48, n= 194 | -2.0736 (60.7226)
  Urate, Year 5, Week 24, n= 184 | -5.296 (65.2308)
  Urate, Year 5, Week 48, n= 178 | -5.7908 (65.6118)
  Urate, Year 6, Week 24, n= 175 | -2.084 (73.3489)
  Urate, Year 6, Week 48, n= 134 | -8.7672 (74.9078)
  Urate, Year 7, Week 24, n= 123 | -2.0775 (72.282)
  Urate, Year 7, Week 48, n= 97 | -0.1021 (60.8139)
  Urate, Year 8, Week 24, n= 60 | 2.0387 (66.4246)
  Urate, Year 8, Week 48, n= 28 | 1.1266 (62.7192)
  Urate, Year 9, Week 24, n= 2 | -1.782 (16.402)
  Urate, Exit, n= 235 | -7.3728 (71.4811)
  Urate, 8 Week, Follow-Up, n= 107 | -6.6934 (84.8414)
  Bilirubin, Year 1, Week 4, n= 251 | 0.008 (2.0889)
  Bilirubin, Year 1, Week 12, n= 248 | 0.165 (2.4872)
  Bilirubin, Year 1, Week 24, n= 246 | 0.075 (2.2546)
  Bilirubin, Year 1, Week 36, n= 238 | 0.124 (2.4316)
  Bilirubin, Year 1, Week 48, n= 250 | 0.231 (2.3675)
  Bilirubin, Year 2, Week 24, n= 248 | 0.359 (2.7306)
  Bilirubin, Year 2, Week 48, n= 233 | 0.307 (3.0385)
  Bilirubin, Year 3, Week 24, n= 218 | 0.249 (2.8298)
  Bilirubin, Year 3, Week 48, n= 209 | -0.115 (2.548)
  Bilirubin, Year 4, Week 24, n= 207 | -0.276 (2.6718)
  Bilirubin, Year 4, Week 48, n= 194 | -0.156 (2.823)
  Bilirubin, Year 5, Week 24, n= 184 | -0.147 (2.8668)
  Bilirubin, Year 5, Week 48, n= 178 | 0.13 (2.7449)
  Bilirubin, Year 6, Week 24, n= 175 | -0.067 (2.7954)
  Bilirubin, Year 6, Week 48, n= 134 | 0.268 (2.6834)
  Bilirubin, Year 7, Week 24, n= 123 | -0.071 (2.7018)
  Bilirubin, Year 7, Week 48, n= 97 | 0.285 (2.85)
  Bilirubin, Year 8, Week 24, n= 60 | 0.529 (2.8249)
  Bilirubin, Year 8, Week 48, n= 28 | 0.175 (2.4435)
  Bilirubin, Year 9, Week 24, n= 2 | -0.45 (1.4142)
  Bilirubin, Exit, n= 235 | 0.403 (2.8268)
  Bilirubin, 8 Week, Follow-Up, n= 107 | -0.191 (3.2759)

12. Primary Outcome: Change From Baseline in Creatinine Clearance at the Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline (BL) (Day 0), at Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion). Change from Baseline in creatinine clearance is summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post- Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Milliliters per second
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Milliliters per second
  Creatinine clearance, Year 1, Week 4, n= 251 | -0.022 (0.2312)
  Creatinine clearance, Year 1, Week 12, n= 248 | 0.01 (0.2455)
  Creatinine clearance, Year 1, Week 24, n= 246 | 0.028 (0.2831)
  Creatinine clearance, Year 1, Week 36, n= 238 | 0.034 (0.3083)
  Creatinine clearance, Year 1, Week 48, n= 250 | 0.017 (0.306)
  Creatinine clearance, Year 2, Week 24, n= 248 | 0.047 (0.3145)
  Creatinine clearance, Year 2, Week 48, n= 233 | 0.04 (0.3498)
  Creatinine clearance, Year 3, Week 24, n= 218 | 0.093 (0.38)
  Creatinine clearance, Year 3, Week 48, n= 209 | 0.093 (0.3784)
  Creatinine clearance, Year 4, Week 24, n= 207 | 0.13 (0.3981)
  Creatinine clearance, Year 4, Week 48, n= 194 | 0.084 (0.3628)
  Creatinine clearance, Year 5, Week 24, n= 184 | 0.087 (0.3724)
  Creatinine clearance, Year 5, Week 48, n= 178 | 0.04 (0.3652)
  Creatinine clearance, Year 6, Week 24, n= 175 | 0.035 (0.3971)
  Creatinine clearance, Year 6, Week 48, n= 134 | 0.039 (0.3985)
  Creatinine clearance, Year 7, Week 24, n= 123 | -0.007 (0.4482)
  Creatinine clearance, Year 7, Week 48, n= 97 | 0.005 (0.4424)
  Creatinine clearance, Year 8, Week 24, n= 60 | -0.018 (0.4682)
  Creatinine clearance, Year 8, Week 48, n= 28 | -0.042 (0.2808)
  Creatinine clearance, Year 9, Week 24, n= 2 | -0.083 (0.165)
  Creatinine clearance, Exit, n= 235 | 0.011 (0.3986)
  Creatinine clearance, 8 Week, Follow-Up, n= 106 | 0.036 (0.3467)

13. Primary Outcome: Change From Baseline in BUN/Creatinine at the Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline (BL) (Day 0), at Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion). Change from Baseline in BUN/creatinine is summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post- Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Ratio
  BUN/creatinine, Year 1, Week 4, n= 251 | -0.2 (4.69)
  BUN/creatinine, Year 1, Week 12, n= 248 | -0.5 (4.86)
  BUN/creatinine, Year 1, Week 24, n= 246 | -0.6 (5.31)
  BUN/creatinine, Year 1, Week 36, n= 238 | -0.4 (5.07)
  BUN/creatinine, Year 1, Week 48, n= 250 | -0.2 (5.29)
  BUN/creatinine, Year 2, Week 24, n= 248 | -0.2 (5.76)
  BUN/creatinine, Year 2, Week 48, n= 233 | 0.3 (4.78)
  BUN/creatinine, Year 3, Week 24, n= 218 | 0.8 (5.63)
  BUN/creatinine, Year 3, Week 48, n= 209 | 0.9 (5.61)
  BUN/creatinine, Year 4, Week 24, n= 207 | 1.2 (5.86)
  BUN/creatinine, Year 4, Week 48, n= 194 | 0.9 (6.05)
  BUN/creatinine, Year 5, Week 24, n= 184 | 1 (5.52)
  BUN/creatinine, Year 5, Week 48, n= 178 | 1.2 (6.49)
  BUN/creatinine, Year 6, Week 24, n= 175 | 1.2 (5.79)
  BUN/creatinine, Year 6, Week 48, n= 134 | 1 (6.38)
  BUN/creatinine, Year 7, Week 24, n= 123 | 1.1 (5.75)
  BUN/creatinine, Year 7, Week 48, n= 97 | 0.7 (5.42)
  BUN/creatinine, Year 8, Week 24, n= 60 | 0.8 (5.09)
  BUN/creatinine, Year 8, Week 48, n= 28 | 0.4 (5.28)
  BUN/creatinine, Year 9, Week 24, n= 2 | -0.5 (0.71)
  BUN/creatinine, Exit, n= 235 | 1.1 (5.57)
  BUN/creatinine, 8 Week, Follow-Up, n= 107 | 1.3 (5.99)

14. Primary Outcome: Change From Baseline in Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Gamma Glutamyl Transferase and Lactate Dehydrogenase at the Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline (BL) (Day 0), at Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 432 weeks and at exit visit. Change from Baseline in alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, gamma glutamyl transferase and lactate dehydrogenase is summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post- Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 432
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Units per liter
  Alanine aminotransferase, Year 1, Week 4, n= 251 | 0.5 (14.89)
  Alanine aminotransferase, Year 1, Week 12, n= 248 | -0.5 (11.01)
  Alanine aminotransferase, Year 1, Week 24, n= 246 | -0.1 (12.27)
  Alanine aminotransferase, Year 1, Week 36, n= 238 | 0.3 (14.12)
  Alanine aminotransferase, Year 1, Week 48, n= 250 | 0.4 (14.64)
  Alanine aminotransferase, Year 2, Week 24, n= 248 | 0.8 (12.33)
  Alanine aminotransferase, Year 2, Week 48, n= 233 | 1.7 (16.67)
  Alanine aminotransferase, Year 3, Week 24, n= 218 | 0.9 (12.32)
  Alanine aminotransferase, Year 3, Week 48, n= 209 | 0.4 (14.93)
  Alanine aminotransferase, Year 4, Week 24, n= 207 | 1.7 (17.02)
  Alanine aminotransferase, Year 4, Week 48, n= 194 | 2.4 (24.4)
  Alanine aminotransferase, Year 5, Week 24, n= 184 | 1.8 (15.79)
  Alanine aminotransferase, Year 5, Week 48, n= 178 | 0.3 (17.15)
  Alanine aminotransferase, Year 6, Week 24, n= 175 | 1 (20.87)
  Alanine aminotransferase, Year 6, Week 48, n= 134 | -0.1 (13.25)
  Alanine aminotransferase, Year 7, Week 24, n= 123 | -2.8 (13.96)
  Alanine aminotransferase, Year 7, Week 48, n= 97 | -2.8 (15.06)
  Alanine aminotransferase, Year 8, Week 24, n= 60 | -5.1 (12.06)
  Alanine aminotransferase, Year 8, Week 48, n= 28 | -0.6 (11.39)
  Alanine aminotransferase, Year 9, Week 24, n= 2 | 5 (4.24)
  Alanine aminotransferase, Exit, n= 235 | -1.2 (13.77)
  Alanine aminotransferase, 8 Week, Follow-Up, n= 10 | 0.1 (14.46)
  Alkaline phosphatase, Year 1, Week 4, n= 251 | -0.8 (13.82)
  Alkaline phosphatase, Year 1, Week 12, n= 248 | 0.4 (17.41)
  Alkaline phosphatase, Year 1, Week 24, n= 246 | 0.3 (16.72)
  Alkaline phosphatase, Year 1, Week 36, n= 238 | 1.2 (16.2)
  Alkaline phosphatase, Year 1, Week 48, n= 250 | 3.3 (19.97)
  Alkaline phosphatase, Year 2, Week 24, n= 248 | 4.9 (21.17)
  Alkaline phosphatase, Year 2, Week 48, n= 233 | 5.8 (21.25)
  Alkaline phosphatase, Year 3, Week 24, n= 218 | 5.4 (20.61)
  Alkaline phosphatase, Year 3, Week 48, n= 209 | 3.1 (21.89)
  Alkaline phosphatase, Year 4, Week 24, n= 207 | 6.5 (29.67)
  Alkaline phosphatase, Year 4, Week 48, n= 194 | 6.2 (33.31)
  Alkaline phosphatase, Year 5, Week 24, n= 184 | 7.8 (24.75)
  Alkaline phosphatase, Year 5, Week 48, n= 178 | 6.7 (26.55)
  Alkaline phosphatase, Year 6, Week 24, n= 175 | 7.5 (33.87)
  Alkaline phosphatase, Year 6, Week 48, n= 134 | 6.6 (26.36)
  Alkaline phosphatase, Year 7, Week 24, n= 123 | 5.5 (25)
  Alkaline phosphatase, Year 7, Week 48, n= 97 | 5.2 (24.83)
  Alkaline phosphatase, Year 8, Week 24, n= 60 | 2.3 (29.63)
  Alkaline phosphatase, Year 8, Week 48, n= 28 | 0.3 (38.97)
  Alkaline phosphatase, Year 9, Week 24, n= 2 | 19.5 (24.75)
  Alkaline phosphatase, Exit, n= 235 | 4.6 (23.59)
  Alkaline phosphatase, 8 Week, Follow-Up, n= 107 | 2.8 (26.98)
  Aspartate aminotransferase ,Year 1, Week 4, n= 242 | 0.3 (11.18)
  Aspartate aminotransferase ,Year 1,Week 12, n= 245 | -0.6 (9.37)
  Aspartate aminotransferase ,Year 1,Week 24, n= 244 | -0.8 (8.14)
  Aspartate aminotransferase,Year 1,Week 36,n=234 | -0.3 (11.29)
  Aspartate aminotransferase ,Year 1,Week 48, n= 250 | -0.2 (10.67)
  Aspartate aminotransferase , Year 2, Week 24,n=246 | 0.4 (10.97)
  Aspartate aminotransferase , Year 2, Week 48,n=231 | 1 (12.24)
  Aspartate aminotransferase , Year 3,Week 24,n=215 | 0.2 (9.49)
  Aspartate aminotransferase ,Year 3,Week 48, n= 205 | 0.1 (14.63)
  Aspartate aminotransferase , Year 4,Week 24, n=204 | 1.3 (14.74)
  Aspartate aminotransferase , Year 4, Week 48,n=191 | 3.7 (32.99)
  Aspartate aminotransferase , Year 5,Week 24, n=184 | 1.7 (16.27)
  Aspartate aminotransferase , Year 5,Week 48, n=176 | 0.6 (15.15)
  Aspartate aminotransferase , Year 6,Week 24,n= 172 | 2.4 (22.03)
  Aspartate aminotransferase , Year 6,Week 48, n=134 | 1 (13.55)
  Aspartate aminotransferase , Year 7,Week 24,n=121 | -0.6 (13.14)
  Aspartate aminotransferase , Year 7, Week 48, n=97 | -1.1 (14.1)
  Aspartate aminotransferase , Year 8, Week 24,n=60 | -2.7 (9.66)
  Aspartate aminotransferase , Year 8, Week 48, n=28 | 0.1 (8.02)
  Aspartate aminotransferase , Year 9, Week 24, n= 2 | 5 (4.24)
  Aspartate aminotransferase , Exit, n= 235 | -0.4 (15.07)
  Aspartate aminotransferase,8 Week,Follow-Up, n=107 | -0.7 (12.45)
  Gamma glutamyl transferase, Year 1, Week 4, n= 251 | 0.5 (22.54)
  Gamma glutamyl transferase, Year 1,Week 12, n= 248 | 0.5 (21.44)
  Gamma glutamyl transferase, Year 1,Week 24, n= 246 | -1.3 (20.21)
  Gamma glutamyl transferase, Year 1, Week 36, n=238 | -0.1 (18.64)
  Gamma glutamyl transferase, Year 1, Week 48, n=250 | 2.2 (39.98)
  Gamma glutamyl transferase, Year 2,Week 24, n= 248 | 1.2 (27.97)
  Gamma glutamyl transferase, Year 2, Week 48,n= 233 | 1.9 (28.88)
  Gamma glutamyl transferase, Year 3, Week 24, n=218 | 1.8 (20.1)
  Gamma glutamyl transferase, Year 3, Week 48, n=209 | -2.4 (31.27)
  Gamma glutamyl transferase, Year 4, Week 24, n=207 | 2.5 (45.58)
  Gamma glutamyl transferase, Year 4, Week 48, n=194 | 1.5 (47.03)
  Gamma glutamyl transferase, Year 5,Week 24, n= 184 | -0.4 (32.51)
  Gamma glutamyl transferase, Year 5, Week 48, n=178 | 0.6 (40.11)
  Gamma glutamyl transferase, Year 6, Week 24, n=175 | -3.3 (40.3)
  Gamma glutamyl transferase, Year 6, Week 48, n=134 | -4.4 (37.08)
  Gamma glutamyl transferase, Year 7, Week 24, n=123 | -7.2 (38.88)
  Gamma glutamyl transferase, Year 7, Week 48, n= 97 | -8.8 (36.19)
  Gamma glutamyl transferase, Year 8, Week 24, n= 60 | -12.9 (35.44)
  Gamma glutamyl transferase, Year 8, Week 48, n= 28 | -6.9 (31.02)
  Gamma glutamyl transferase, Year 9, Week 24, n= 2 | 2.5 (3.54)
  Gamma glutamyl transferase, Exit, n= 235 | -2.2 (35.29)
  Gamma glutamyl transferase, 8 Week,Follow-Up,n=107 | 2.1 (35.9)
  Lactate dehydrogenase , Year 1, Week 4, n= 242 | 0.2 (26.46)
  Lactate dehydrogenase , Year 1, Week 12, n= 245 | -2.4 (29.56)
  Lactate dehydrogenase , Year 1, Week 24, n= 244 | -2.2 (37.57)
  Lactate dehydrogenase , Year 1, Week 36, n= 234 | -2.8 (34.88)
  Lactate dehydrogenase , Year 1, Week 48, n= 250 | -4.3 (35.5)
  Lactate dehydrogenase , Year 2, Week 24, n= 246 | -4.8 (36.29)
  Lactate dehydrogenase , Year 2, Week 48, n= 231 | -5.4 (40.42)
  Lactate dehydrogenase , Year 3, Week 24, n= 215 | -8.1 (40.13)
  Lactate dehydrogenase , Year 3, Week 48, n= 205 | -9.2 (47.95)
  Lactate dehydrogenase , Year 4, Week 24, n= 204 | -7.7 (45.12)
  Lactate dehydrogenase , Year 4, Week 48, n= 191 | -4.7 (53.17)
  Lactate dehydrogenase , Year 5, Week 24, n= 184 | -5.5 (48.34)
  Lactate dehydrogenase , Year 5, Week 48, n= 176 | -10.3 (49.81)
  Lactate dehydrogenase , Year 6, Week 24, n= 172 | -2.7 (72.28)
  Lactate dehydrogenase , Year 6, Week 48, n= 134 | -5.3 (55.64)
  Lactate dehydrogenase , Year 7, Week 24, n= 121 | -7.9 (53.17)
  Lactate dehydrogenase , Year 7, Week 48, n= 97 | -9.5 (57.15)
  Lactate dehydrogenase , Year 8, Week 24, n= 60 | -11.2 (58.81)
  Lactate dehydrogenase , Year 8, Week 48, n= 28 | -5.5 (81.78)
  Lactate dehydrogenase , Year 9, Week 24, n= 2 | -9.5 (0.71)
  Lactate dehydrogenase , Exit, n= 235 | -6.5 (56.73)
  Lactate dehydrogenase , 8 Week, Follow-Up, n= 107 | -3.4 (52.66)

15. Primary Outcome: Number of Participants With the Indicated Immunogenic Response
Description: Immunogenic response was assessed by binding confirmatory assay at Baseline (BL) (Day 0), at Week 24 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion). Number of participants with the indicated immunogenic response are summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Results of binding confirmatory assay were categorized as negative, persistent positive (defined as a positive immunogenic response that occurs at least 2 consecutive assessments or a single result at the final assessment) or transient positive (defined as a single positive immunogenic response that does not occur at the final assessment). Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Participants
  Negative, Year 0-1, n=267 | 262
  Negative, Year 1-2, n=255 | 251
  Negative, Year 2-3, n=240 | 239
  Negative, Year 3-4, n=214 | 213
  Negative, Year 4-5, n=195 | 195
  Negative, Year 5-6, n=185 | 185
  Negative, Year 6-7, n=125 | 125
  Negative, Year 7 plus, n=63 | 63
  Transient positive, Year 0-1, n=267 | 5
  Transient positive, Year 1-2, n=255 | 4
  Transient positive, Year 2-3, n=240 | 0
  Transient positive, Year 3-4, n=214 | 1
  Transient positive, Year 4-5, n=195 | 0
  Transient positive, Year 5-6, n=185 | 0
  Transient positive, Year 6-7, n=125 | 0
  Transient positive, Year 7 plus, n=63 | 0
  Persistent positive, Year 0-1, n=267 | 0
  Persistent positive, Year 1-2, n=255 | 0
  Persistent positive, Year 2-3, n=240 | 0
  Persistent positive, Year 3-4, n=214 | 0
  Persistent positive, Year 4-5, n=195 | 0
  Persistent positive, Year 5-6, n=185 | 0
  Persistent positive, Year 6-7, n=125 | 0
  Persistent positive, Year 7 plus, n=63 | 0
  Unknown, Year 0-1, n=267 | 0
  Unknown, Year 1-2, n=255 | 0
  Unknown, Year 2-3, n=240 | 1
  Unknown, Year 3-4, n=214 | 0
  Unknown, Year 4-5, n=195 | 0
  Unknown, Year 5-6, n=185 | 0
  Unknown, Year 6-7, n=125 | 0
  Unknown, Year 7 plus, n=63 | 0

16. Primary Outcome: Systolic Blood Pressure and Diastolic Blood Pressure at Indicated Time Points.
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) was measured at Baseline (BL) (Day 0), at Week 24 and 48 in first year, at Week 24 and 48 in subsequent years up to 432 weeks and at exit visit. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 432
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Millimeters of mercury
  DBP, Baseline, n= 268 | 74.3 (9.92)
  DBP, Year 1 , Week 24, n= 255 | 74.5 (9.96)
  DBP, Year 1 , Week 48, n= 255 | 73.5 (9.92)
  DBP, Year 2 , Week 24, n= 251 | 74.5 (11.01)
  DBP, Year 2 , Week 48, n= 236 | 73.5 (10.17)
  DBP, Year 3 , Week 24, n= 223 | 73.6 (10.32)
  DBP, Year 3 , Week 48, n= 214 | 73.4 (10.12)
  DBP, Year 4 , Week 24, n= 214 | 74.4 (9.56)
  DBP, Year 4 , Week 48, n= 199 | 75.2 (10.52)
  DBP, Year 5 , Week 24, n= 187 | 74.3 (9.89)
  DBP, Year 5 , Week 48, n= 185 | 73.4 (10.15)
  DBP, Year 6 , Week 24, n= 178 | 74.1 (10.25)
  DBP, Year 6 , Week 48, n= 138 | 73.9 (10.78)
  DBP, Year 7 , Week 24, n= 124 | 75.2 (9.5)
  DBP, Year 7 , Week 48, n= 98 | 73.1 (9.94)
  DBP, Year 8 , Week 24, n= 60 | 73.4 (9.79)
  DBP, Year 8 , Week 48, n= 29 | 73.6 (8.27)
  DBP, Year 9 , Week 24, n= 2 | 90 (12.73)
  DBP, Exit, n= 233 | 75.2 (9.77)
  SBP, Baseline, n= 268 | 119.7 (15.75)
  SBP, Year 1 , Week 24, n= 255 | 120 (16.14)
  SBP, Year 1 , Week 48, n= 255 | 120.2 (14.66)
  SBP, Year 2 , Week 24, n= 251 | 120.1 (16.49)
  SBP, Year 2 , Week 48, n= 236 | 119.1 (15.22)
  SBP, Year 3 , Week 24, n= 223 | 120.7 (16.23)
  SBP, Year 3 , Week 48, n= 214 | 120.2 (14.44)
  SBP, Year 4 , Week 24, n= 214 | 121.4 (14.61)
  SBP, Year 4 , Week 48, n= 199 | 121.4 (15.03)
  SBP, Year 5 , Week 24, n= 187 | 120.7 (14.92)
  SBP, Year 5 , Week 48, n= 185 | 119.9 (15.29)
  SBP, Year 6 , Week 24, n= 178 | 121.5 (15.29)
  SBP, Year 6 , Week 48, n= 138 | 121.7 (15.86)
  SBP, Year 7 , Week 24, n= 124 | 121.6 (14.73)
  SBP, Year 7 , Week 48, n= 98 | 120.6 (14.19)
  SBP, Year 8 , Week 24, n= 60 | 120.5 (14.65)
  SBP, Year 8 , Week 48, n= 29 | 118.2 (11.73)
  SBP, Year 9 , Week 24, n= 2 | 115.5 (6.36)
  SBP, Exit, n= 233 | 123.3 (15.53)

17. Primary Outcome: Percentage of Participants With at Least 25% Increase From Baseline in Creatinine at Indicated Time Points.
Description: Serum creatinine was assessed at Baseline (BL) (Day 0), at Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion). Percentage of participants with at least 25% increase from baseline in creatinine are summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Number; unit: Percentage of Participants
Groups:
- Belimumab 10 mg/kg IV (Placebo): Participants, who had received placebo in study HGS1006-C1056, received intravenous (IV) infusion of belimumab 10 mg/kg body weight over 1 hour every 28 days. The first dose of belimumab was given 4 weeks (2 to 8 weeks) after the last dose in the HGS1006-C1056 study. The dosing was continued for five years from the time the last participant enrolled in the study or until there were 100 or fewer participants enrolled. All participants received standard of care (SoC) for systemic lupus erythematosus (SLE) during study participation.
- Belimumab 10 mg/kg IV (Belimumab): Participants, who had received belimumab 1mg/kg or 10 mg/kg in study HGS1006-C1056, received intravenous (IV) infusion of belimumab 10 mg/kg body weight over 1 hour every 28 days. The first dose of belimumab was given 4 weeks (2 to 8 weeks) after the last dose in the HGS1006-C1056 study. The dosing was continued for five years from the time the last participant enrolled in the study or until there were 100 or fewer participants enrolled. All participants received standard of care (SoC) for systemic lupus erythematosus (SLE) during study participation.
Arm/Group | Belimumab 10 mg/kg IV (Placebo) | Belimumab 10 mg/kg IV (Belimumab)
Number analyzed (Participants) | 91 | 177
Percentage of Participants
  Year 0-1, n= 91, 177 | 7.7 | 23.2
  Year 1-2, n= 79, 177 | 3.8 | 20.3
  Year 2-3, n= 75, 168 | 2.7 | 8.3
  Year 3-4, n= 68, 150 | 4.4 | 6
  Year 4-5, n= 61, 139 | 4.9 | 9.4
  Year 5-6, n= 59, 132 | 5.1 | 9.1
  Year 6-7, n= 12, 118 | 8.3 | 11.9
  Year 7+, n= 0, 65 | 0 | 10.8

18. Primary Outcome: Percentage of Participants With at Least 25% Reduction From Baseline in Creatinine at Indicated Time Points. Amongst Subjects With Abnormal (>124 Umol/L) Creatinine at Baseline by Year Interval.
Description: Serum creatinine was assessed at Baseline (BL) (Day 0), at Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion). Percentage of participants with at least 25% reduction from baseline in creatinine are summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population. Only those subjects with abnormal (>124 umol/L) creatinine at baseline by year interval.
Measure: Number; unit: Percentage of Participants
Arm/Group | Belimumab 10 mg/kg IV (Placebo) | Belimumab 10 mg/kg IV (Belimumab)
Number analyzed (Participants) | 91 | 177
Percentage of Participants
  Year 0-1, n= 6, 3 | 16.7 | 33.3
  Year 1-2, n= 5, 3 | 20 | 0
  Year 2-3, n= 3, 3 | 33.3 | 0
  Year 3-4, n= 2, 2 | 0 | 50
  Year 4-5, n= 2, 2 | 0 | 50
  Year 5-6, n= 2, 2 | 50 | 0
  Year 6-7, n= 1, 1 | 0 | 100
  Year 7+, n= 0, 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Serum Immunoglobulins Below the Lower Limit of Normal at Indicated Time Points.
Description: Serum immunoglobulin G (IgG) was collected at Baseline (BL) (Day 0), at Week 24 and Week 48 in first year, at Week 48 in subsequent years up to 8 years and at follow-up (up to 8 weeks post last infusion). Number of participants with serum immunoglobulins below the lower limit of normal (LLN) (<0.5 nanograms per milliliter [ng/mL]) are summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 392
Population: MITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Participants
  Baseline, n=268 | 8
  Year 1, Week 24, n= 252 | 14
  Year 1, Week 48, n= 255 | 16
  Year 2, Week 48, n= 237 | 19
  Year 3, Week 48, n= 224 | 17
  Year 4, Week 48, n= 208 | 26
  Year 5, Week 48, n= 190 | 19
  Year 6, Week 48, n= 150 | 21
  Year 7, Week 48, n= 112 | 21
  Year 8, Week 48, n= 59 | 5
  Exit, n= 235 | 29
  8 Week Follow-Up, n= 106 | 10

20. Secondary Outcome: Percentage of Participants Achieving SRI Response at Indicated Time Points
Description: The percentage of participants achieving a SLE Responder Index (SRI) response at Baseline (BL) (Day 0), at Week 4, 12, 24, 36 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at follow-up (up to 8 weeks post last infusion) are summarized. The BL is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Response is defined as:>=4 point reduction from the BL in the safety of estrogen in lupus national assessment (SELENA) SLE disease activity index (SLEDAI) score and no worsening (increase of <0.30 points from the BL) in Physicians Global Assessment (PGA), and no new British Isles Lupus Assessment Group (BILAG) A organ domain score or 2 new BILAG B organ domain scores compared with the BL. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MIIT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Percentage of Participants
  Year 1 , Week 24, n= 229 | 41.9
  Year 1 , Week 48, n= 225 | 45.3
  Year 2 , Week 24, n= 227 | 49.3
  Year 2 , Week 48, n= 204 | 49
  Year 3 , Week 24, n= 211 | 51.2
  Year 3 , Week 48, n= 185 | 58.4
  Year 4 , Week 24, n= 188 | 56.9
  Year 4 , Week 48, n= 174 | 64.9
  Year 5 , Week 24, n= 168 | 66.7
  Year 5 , Week 48, n= 157 | 62.4
  Year 6 , Week 24, n= 164 | 69.5
  Year 6 , Week 48, n= 123 | 74
  Year 7 , Week 24, n= 119 | 75.6
  Year 7 , Week 48, n= 93 | 78.5
  Year 8 , Week 24, n= 63 | 66.7
  Year 8 , Week 48, n= 29 | 65.5
  Year 9 , Week 24, n= 2 | 0

21. Secondary Outcome: Observed Anti-double Stranded DNA Levels at Indicated Time Points.
Description: Anti-double stranded deoxyribonucleic acid (anti-dsDNA) levels were assessed at Baseline (BL) (Day 0), at Week 24 and 48 in first year, at Week 24 and 48 in subsequent years up to 432 weeks in participants who were positive at baseline (anti-dsDNA >=30 International Units/milliliter [IU/mL]). Observed anti-dsDNA levels are summarized. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 432
Population: MITT Population
Measure: Median (Full Range); unit: International units per milliliter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 135
International units per milliliter
  Baseline, n= 135 | 193 [34 to 201]
  Year 1, Week 24, n= 128 | 127.5 [29 to 201]
  Year 1, Week 48, n= 130 | 123 [29 to 201]
  Year 2, Week 24, n= 126 | 93.5 [29 to 349]
  Year 2, Week 48, n= 128 | 95 [5 to 2505]
  Year 3, Week 24, n= 120 | 82.5 [5 to 1545]
  Year 3, Week 48, n= 116 | 86.5 [5 to 556]
  Year 4, Week 24, n= 112 | 87.5 [5 to 2305]
  Year 4, Week 48, n= 100 | 76.5 [5 to 1873]
  Year 5, Week 24, n= 98 | 60 [5 to 1188]
  Year 5, Week 48, n= 96 | 47.5 [5 to 1765]
  Year 6, Week 24, n= 87 | 47 [5 to 1863]
  Year 6, Week 48, n= 66 | 50 [5 to 1018]
  Year 7, Week 24, n= 63 | 35 [5 to 2648]
  Year 7, Week 48, n= 48 | 32 [5 to 736]
  Year 8, Week 24, n= 35 | 29 [5 to 521]
  Year 8, Week 48, n= 16 | 50.5 [5 to 439]
  Year 9, Week 24, n= 1 | 45 [45 to 45]
  Exit, n= 120 | 37 [5 to 1608]

22. Secondary Outcome: Median Percent Change From Baseline in Anti-double Stranded DNA at Indicated Time Points.
Description: Anti-dsDNA levels were assessed at Baseline (BL) (Day 0), 24 and 48 in first year, at Week 24 and 48 in subsequent years up to 432 weeks and at exit visit in participants who were positive at baseline (anti-dsDNA ≥30 IU/mL). Median percent change from Baseline in anti-dsDNA levels are summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Percent change from Baseline is calculated as: 100 x ([Post-Dose Visit Value - Baseline] / Baseline). Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 432
Population: MITT Population
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 135
Percentage change
  Year 1, Week 24, n= 128 | -9.77 [-75.6 to 54.6]
  Year 1, Week 48, n= 130 | -15.58 [-84.2 to 183.1]
  Year 2, Week 24, n= 126 | -27.5 [-84.7 to 181.7]
  Year 2, Week 48, n= 128 | -30.12 [-90.6 to 1253.6]
  Year 3, Week 24, n= 120 | -34.22 [-90.6 to 668.7]
  Year 3, Week 48, n= 116 | -34.92 [-90.6 to 176.6]
  Year 4, Week 24, n= 112 | -38.58 [-90.6 to 1046.8]
  Year 4, Week 48, n= 100 | -54.46 [-96 to 831.8]
  Year 5, Week 24, n= 98 | -54.39 [-96.5 to 491]
  Year 5, Week 48, n= 96 | -64.43 [-97.5 to 778.1]
  Year 6, Week 24, n= 87 | -64.04 [-97.5 to 826.9]
  Year 6, Week 48, n= 66 | -64.91 [-97.5 to 406.5]
  Year 7, Week 24, n= 63 | -74.74 [-97.5 to 1217.4]
  Year 7, Week 48, n= 48 | -78.15 [-97.5 to 557.1]
  Year 8, Week 24, n= 35 | -79.1 [-97.5 to 365.2]
  Year 8, Week 48, n= 16 | -72.38 [-97.5 to 292]
  Year 9, Week 24, n= 1 | -77.6 [-77.6 to -77.6]
  Exit, n= 120 | -66.67 [-97.5 to 700]

23. Secondary Outcome: Observed Complement C3 and C4 Levels at Indicated Time Points
Description: Complement C3 and C4 levels were assessed at Baseline (BL) (Day 0), at Week 24 and 48 in first year, at Week 24 and 48 in subsequent years up to 440 weeks and at exit visit in participants with low complements at Baseline (C3 <90 milligram per deciliter (mg/dL) and C4 <16 mg/dL). Observed complement C3 and C4 levels are summarized. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 440
Population: MITT Population
Measure: Median (Full Range); unit: Milligrams per deciliter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 135
Milligrams per deciliter
  C3, Baseline, n= 86 | 76 [40 to 89]
  C3, Year 1, Week 24, n= 83 | 80 [43 to 160]
  C3, Year 1, Week 48, n= 83 | 86 [38 to 144]
  C3, Year 2, Week 24, n= 81 | 85 [46 to 157]
  C3, Year 2, Week 48, n= 80 | 88.5 [36 to 137]
  C3, Year 3, Week 24, n= 74 | 90.5 [55 to 133]
  C3, Year 3, Week 48, n= 73 | 93 [51 to 139]
  C3, Year 4, Week 24, n= 72 | 94 [47 to 150]
  C3, Year 4, Week 48, n= 66 | 95 [58 to 137]
  C3, Year 5, Week 24, n= 63 | 99 [64 to 193]
  C3, Year 5, Week 48, n= 61 | 97 [56 to 172]
  C3, Year 6, Week 24, n= 55 | 99 [54 to 161]
  C3, Year 6, Week 48, n= 37 | 103 [47 to 158]
  C3, Year 7, Week 24, n= 41 | 103 [50 to 147]
  C3, Year 7, Week 48, n= 32 | 110 [51 to 173]
  C3, Year 8, Week 24, n= 20 | 110.5 [76 to 177]
  C3, Year 8, Week 48, n= 9 | 104 [79 to 158]
  C3, Exit, n= 74 | 103 [56 to 173]
  C4, Baseline, n=98 | 10 [3 to 15]
  C4, Year 1, Week 24, n=95 | 13 [3 to 25]
  C4, Year 1, Week 48, n=93 | 15 [4 to 28]
  C4, Year 2, Week 24, n=93 | 15 [3 to 29]
  C4, Year 2, Week 48, n=94 | 16 [4 to 37]
  C4, Year 3, Week 24, n=84 | 15.5 [4 to 31]
  C4, Year 3, Week 48, n=83 | 16 [3 to 35]
  C4, Year 4, Week 24, n=81 | 16 [3 to 38]
  C4, Year 4, Week 48, n=71 | 17 [4 to 26]
  C4, Year 5, Week 24, n=70 | 18 [4 to 40]
  C4, Year 5, Week 48, n=70 | 18 [3 to 39]
  C4, Year 6, Week 24, n=62 | 18 [5 to 36]
  C4, Year 6, Week 48, n=45 | 18 [5 to 29]
  C4, Year 7, Week 24, n=49 | 19 [6 to 34]
  C4, Year 7, Week 48, n=35 | 19 [6 to 34]
  C4, Year 8, Week 24, n=24 | 20.5 [10 to 35]
  C4, Year 8, Week 48, n=12 | 18 [7 to 36]
  C4, Year 9, Week 24, n=1 | 22 [22 to 22]
  C4, Exit, n=85 | 18 [4 to 41]

24. Secondary Outcome: Median Percent Change From Baseline in Complement C3 and C4 Levels at Indicated Time Points
Description: Complement C3 and C4 levels were assessed at Baseline (BL) (Day 0), 24 and 48 in first year, at Week 24 and 48 in subsequent years up to 432 weeks and at exit visit in participants with low complements at Baseline (C3 <90 milligrams per decilitre (mg/dL) and C4 <16 mg/dL). Median percent change from Baseline in complement C3 and C4 levels are summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Percent change from Baseline is calculated as: 100 x ([Post-Dose Visit Value - Baseline] / Baseline). Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 432
Population: MITT Population
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 135
Percent Change
  C3, Year 1, Week 24, n= 83 | 10.91 [-33 to 281]
  C3, Year 1, Week 48, n= 83 | 17.86 [-45.3 to 104.8]
  C3, Year 2, Week 24, n= 81 | 18.64 [-23.3 to 192.9]
  C3, Year 2, Week 48, n= 80 | 16.71 [-37.9 to 163.3]
  C3, Year 3, Week 24, n= 74 | 24.26 [-17.3 to 161.2]
  C3, Year 3, Week 48, n= 73 | 22.73 [-34.6 to 163.3]
  C3, Year 4, Week 24, n= 72 | 32.43 [-32.9 to 206.1]
  C3, Year 4, Week 48, n= 66 | 30.63 [-27.5 to 177.6]
  C3, Year 5, Week 24, n= 63 | 33.93 [-24.7 to 175.7]
  C3, Year 5, Week 48, n= 61 | 34.29 [-17.9 to 173.5]
  C3, Year 6, Week 24, n= 55 | 35.71 [-18 to 159.7]
  C3, Year 6, Week 48, n= 37 | 34.57 [-32.9 to 166.7]
  C3, Year 7, Week 24, n= 41 | 36.11 [-34.2 to 137.1]
  C3, Year 7, Week 48, n= 32 | 42.04 [-36.3 to 179]
  C3, Year 8, Week 24, n= 20 | 36.97 [7.7 to 185.5]
  C3, Year 8, Week 48, n= 9 | 30.16 [5 to 163.3]
  C3, Exit, n= 74 | 39.05 [-25.6 to 195.2]
  C4, Year 1, Week 24, n=95 | 30.77 [-53.3 to 275]
  C4, Year 1, Week 48, n=93 | 40 [-40 to 200]
  C4, Year 2, Week 24, n=93 | 42.86 [-57.1 to 350]
  C4, Year 2, Week 48, n=94 | 47.73 [-33.3 to 270]
  C4, Year 3, Week 24, n=84 | 50 [-20 to 266.7]
  C4, Year 3, Week 48, n=83 | 46.15 [-40 to 250]
  C4, Year 4, Week 24, n=81 | 57.14 [-70 to 450]
  C4, Year 4, Week 48, n=71 | 58.33 [-42.9 to 433.3]
  C4, Year 5, Week 24, n=70 | 70.33 [-30 to 500]
  C4, Year 5, Week 48, n=70 | 65.15 [-40 to 566.7]
  C4, Year 6, Week 24, n=62 | 71.36 [-10 to 800]
  C4, Year 6, Week 48, n=45 | 57.14 [-40 to 600]
  C4, Year 7, Week 24, n=49 | 63.64 [-40 to 700]
  C4, Year 7, Week 48, n=35 | 62.5 [-14.3 to 900]
  C4, Year 8, Week 24, n=24 | 78.97 [0 to 900]
  C4, Year 8, Week 48, n=12 | 69.74 [-30 to 1100]
  C4, Year 9, Week 24, n=1 | 100 [100 to 100]
  C4, Exit, n=85 | 75 [-53.8 to 1066.7]

25. Secondary Outcome: Percent of Participants With Daily Prednisone Dose Reduction at Indicated Time Points.
Description: Trends for reduction in prednisone use in participants receiving belimumab were observed up to 432 weeks. Percentage of participants with daily prednisone dose reduced to <=7.5 mg/day from >7.5 mg/kg at the Baseline are summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 432
Population: MITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 86
Percentage of Participants
  Year 1, Week 24, n= 80 | 2.5
  Year 1, Week 48, n= 81 | 21
  Year 2, Week 24, n= 78 | 38.5
  Year 2, Week 48, n= 76 | 40.8
  Year 3, Week 24, n= 64 | 50
  Year 3, Week 48, n= 63 | 41.3
  Year 4, Week 24, n= 65 | 43.1
  Year 4, Week 48, n= 62 | 37.1
  Year 5, Week 24, n= 57 | 33.3
  Year 5, Week 48, n= 57 | 38.6
  Year 6, Week 24, n= 55 | 34.5
  Year 6, Week 48, n= 47 | 42.6
  Year 7, Week 24, n= 42 | 38.1
  Year 7, Week 48, n= 38 | 39.5
  Year 8, Week 24, n= 24 | 50
  Year 8, Week 48, n= 12 | 58.3
  Year 9, Week 24, n= 2 | 100

26. Secondary Outcome: Percent of Participants With >= 50% Reduction in Proteinuria at Indicated Time Points.
Description: Proteinuria is defined as the presence of an excess of serum proteins in the urine. Trends for reduction in proteinuria in participants receiving belimumab were assessed up to 432 weeks and at Exit visit. Percentage of participants with >= 50% reduction in proteinuria among participants with Baseline proteinuria >0.5 g/24 hour (hr) are summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 432
Population: MITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 36
Percentage of Participants
  Year 1, Week 24, n=34 | 41.2
  Year 1, Week 48, n=33 | 63.6
  Year 2, Week 24, n=33 | 60.6
  Year 2, Week 48, n=30 | 53.3
  Year 3, Week 24, n=31 | 74.2
  Year 3, Week 48, n=28 | 67.9
  Year 4, Week 24, n=25 | 88
  Year 4, Week 48, n=23 | 73.9
  Year 5, Week 24, n=23 | 73.9
  Year 5, Week 48, n=22 | 86.4
  Year 6, Week 24, n=22 | 77.3
  Year 6, Week 48, n=17 | 76.5
  Year 7, Week 24, n=14 | 78.6
  Year 7, Week 48, n=7 | 71.4
  Year 8, Week 24, n=4 | 75
  Year 8, Week 48, n=1 | 100
  Year 9, Week 24, n=28 | 64.3

27. Secondary Outcome: Observed B-cell Levels at Indicated Time Points.
Description: B-cell levels were assessed at Baseline (BL) (Day 0), Week (Wk) 24 and 48 in first year, at Week 24 and 48 in subsequent years up to 432 weeks and at exit visit. Observed absolute B cell subsets (CD20+), CD19+/27BRIGHT/38BRIGHT SLE subset, CD19+20-27hi+ short-lived plasma cells (SLPC), CD20+/138+ plasmacytoid, CD20+/27+ memory, CD20+/27- naïve, CD20+/69+activated, CD20-/138+ plasma cells, Total CD19+ B-cells (CD19+) levels are summarized. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 432
Population: MITT Population
Measure: Median (Full Range); unit: Cell count
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Cell count
  CD20+, Baseline, n= 262 | 112.5 [2 to 807]
  CD20+, Yr 1, Wk 24, n= 251 | 68 [2 to 433]
  CD20+, Yr 1, Wk 48, n= 242 | 50 [2 to 407]
  CD20+, Yr 2, Wk 24, n= 238 | 37.5 [5 to 278]
  CD20+, Yr 2, Wk 48, n= 224 | 34 [5 to 1528]
  CD20+, Yr 3, Wk 24, n= 212 | 31 [5 to 293]
  CD20+, Yr 3, Wk 48, n= 202 | 26 [5 to 500]
  CD20+, Yr 4, Wk 24, n= 196 | 27 [3 to 355]
  CD20+, Yr 4, Wk 48, n= 181 | 23 [5 to 238]
  CD20+, Yr 5, Wk 24, n= 172 | 22 [1 to 141]
  CD20+, Yr 5, Wk 48, n= 166 | 18.5 [5 to 248]
  CD20+, Yr 6, Wk 24, n= 159 | 21 [4 to 397]
  CD20+, Yr 6, Wk 48, n= 114 | 20 [4 to 113]
  CD20+, Yr 7, Wk 24, n= 111 | 20 [4 to 158]
  CD20+, Yr 7, Wk 48, n= 87 | 21 [5 to 120]
  CD20+, Yr 8, Wk 24, n= 54 | 17 [5 to 91]
  CD20+, Yr 8, Wk 48, n= 28 | 15.5 [5 to 57]
  CD20+, Yr 9, Wk 24, n= 2 | 7.5 [7 to 8]
  CD20+, Exit, n= 207 | 22 [3 to 364]
  CD19+/27BRIGHT/38BRIGHT SLE, Baseline, n= 262 | 17 [0 to 600]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 1, Wk 24, n= 251 | 13 [0 to 452]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 1, Wk 48, n= 247 | 12 [0 to 177]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 2, Wk 24, n= 246 | 14 [0 to 204]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 2, Wk 48, n= 233 | 13 [0 to 345]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 3, Wk 24, n= 218 | 12 [0 to 216]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 3, Wk 48, n= 212 | 12 [0 to 331]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 4, Wk 24, n= 211 | 14 [0 to 407]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 4, Wk 48, n= 194 | 14 [0 to 442]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 5, Wk 24, n= 189 | 11 [0 to 414]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 5, Wk 48, n= 181 | 11 [0 to 591]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 6, Wk 24, n= 174 | 10.5 [0 to 443]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 6, Wk 48, n= 133 | 10 [0 to 248]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 7, Wk 24, n= 122 | 9 [0 to 381]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 7, Wk 48, n= 97 | 8 [0 to 156]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 8, Wk 24, n= 60 | 6.5 [0 to 755]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 8, Wk 48, n= 29 | 5 [0 to 39]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 9, Wk 24, n= 2 | 17.5 [6 to 29]
  CD19+/27BRIGHT/38BRIGHT SLE, Exit, n= 232 | 9 [0 to 555]
  CD19+20-27hi+ SLPC, Baseline, n= 258 | 16 [0 to 585]
  CD19+20-27hi+ SLPC, Yr 1, Wk 24, n= 247 | 13 [0 to 443]
  CD19+20-27hi+ SLPC, Yr 1, Wk 48, n= 244 | 11 [0 to 145]
  CD19+20-27hi+ SLPC, Yr 2, Wk 24, n= 244 | 13 [0 to 289]
  CD19+20-27hi+ SLPC, Yr 2, Wk 48, n= 233 | 13 [0 to 316]
  CD19+20-27hi+ SLPC, Yr 3, Wk 24, n= 218 | 12 [0 to 210]
  CD19+20-27hi+ SLPC, Yr 3, Wk 48, n= 211 | 12 [0 to 324]
  CD19+20-27hi+ SLPC, Yr 4, Wk 24, n= 210 | 13 [0 to 364]
  CD19+20-27hi+ SLPC, Yr 4, Wk 48, n= 193 | 12 [0 to 452]
  CD19+20-27hi+ SLPC, Yr 5, Wk 24, n= 188 | 10.5 [0 to 377]
  CD19+20-27hi+ SLPC, Yr 5, Wk 48, n= 181 | 10 [0 to 597]
  CD19+20-27hi+ SLPC, Yr 6, Wk 24, n= 174 | 9 [0 to 400]
  CD19+20-27hi+ SLPC, Yr 6, Wk 48, n= 133 | 8 [0 to 227]
  CD19+20-27hi+ SLPC, Yr 7, Wk 24, n= 122 | 9 [0 to 328]
  CD19+20-27hi+ SLPC, Yr 7, Wk 48, n= 97 | 9 [0 to 156]
  CD19+20-27hi+ SLPC, Yr 8, Wk 24, n= 60 | 9 [0 to 754]
  CD19+20-27hi+ SLPC, Yr 8, Wk 48, n= 29 | 4 [0 to 42]
  CD19+20-27hi+ SLPC, Yr 9, Wk 24, n= 2 | 16 [4 to 28]
  CD19+20-27hi+ SLPC, Exit, n= 233 | 9 [0 to 603]
  CD20+/138+ plasmacytoid, Baseline, n= 261 | 95 [0 to 4274]
  CD20+/138+ plasmacytoid, Yr 1, Wk 24, n= 251 | 64 [1 to 1613]
  CD20+/138+ plasmacytoid, Yr 1, Wk 48, n= 247 | 37 [2 to 962]
  CD20+/138+ plasmacytoid, Yr 2, Wk 24, n= 246 | 32.5 [0 to 221]
  CD20+/138+ plasmacytoid, Yr 2, Wk 48, n= 233 | 27 [1 to 249]
  CD20+/138+ plasmacytoid, Yr 3, Wk 24, n= 218 | 24 [0 to 322]
  CD20+/138+ plasmacytoid, Yr 3, Wk 48, n= 212 | 12 [0 to 220]
  CD20+/138+ plasmacytoid, Yr 4, Wk 24, n= 211 | 8 [0 to 128]
  CD20+/138+ plasmacytoid, Yr 4, Wk 48, n= 194 | 5 [0 to 246]
  CD20+/138+ plasmacytoid, Yr 5, Wk 24, n= 189 | 4 [0 to 136]
  CD20+/138+ plasmacytoid, Yr 5, Wk 48, n= 181 | 3 [0 to 102]
  CD20+/138+ plasmacytoid, Yr 6, Wk 24, n= 174 | 3 [0 to 38]
  CD20+/138+ plasmacytoid, Yr 6, Wk 48, n= 133 | 3 [0 to 25]
  CD20+/138+ plasmacytoid, Yr 7, Wk 24, n= 122 | 2 [0 to 70]
  CD20+/138+ plasmacytoid, Yr 7, Wk 48, n= 97 | 2 [0 to 23]
  CD20+/138+ plasmacytoid, Yr 8, Wk 24, n= 60 | 2 [0 to 18]
  CD20+/138+ plasmacytoid, Yr 8, Wk 48, n= 29 | 1 [0 to 16]
  CD20+/138+ plasmacytoid, Yr 9, Wk 24, n= 2 | 1 [0 to 2]
  CD20+/138+ plasmacytoid, Exit, n= 232 | 3 [0 to 231]
  CD20+/27+Memory, Baseline, n= 262 | 17 [0 to 177]
  CD20+/27+Memory, Yr 1, Wk 24, n= 251 | 30 [1 to 279]
  CD20+/27+Memory, Yr 1, Wk 48, n= 242 | 23 [0 to 275]
  CD20+/27+Memory, Yr 2, Wk 24, n= 238 | 17 [1 to 181]
  CD20+/27+Memory, Yr 2, Wk 48, n= 224 | 16 [1 to 686]
  CD20+/27+Memory, Yr 3, Wk 24, n= 212 | 13 [0 to 88]
  CD20+/27+Memory, Yr 3, Wk 48, n= 202 | 11 [1 to 342]
  CD20+/27+Memory, Yr 4, Wk 24, n= 196 | 10.5 [1 to 276]
  CD20+/27+Memory, Yr 4, Wk 48, n= 181 | 9 [1 to 196]
  CD20+/27+Memory, Yr 5, Wk 24, n= 172 | 8.5 [1 to 76]
  CD20+/27+Memory, Yr 5, Wk 48, n= 166 | 7 [1 to 166]
  CD20+/27+Memory, Yr 6,Wk 24,n=158 | 7 [1 to 73]
  CD20+/27+Memory, Yr 6, Wk 48, n= 114 | 6 [1 to 46]
  CD20+/27+Memory, Yr 7, Wk 24, n= 111 | 6 [1 to 91]
  CD20+/27+Memory, Yr 7, Wk 48, n= 87 | 6 [1 to 81]
  CD20+/27+Memory, Yr 8, Wk 24, n= 54 | 5 [1 to 34]
  CD20+/27+Memory, Yr 8, Wk 48, n= 28 | 6 [1 to 32]
  CD20+/27+Memory, Yr 9, Wk 24, n= 2 | 2 [1 to 3]
  CD20+/27+Memory, Exit, n= 207 | 8 [0 to 167]
  CD20+/27-naive, Baseline, n= 262 | 88 [1 to 717]
  CD20+/27-naive, Yr 1, Wk 24, n= 251 | 36 [1 to 371]
  CD20+/27-naive, Yr 1, Wk 48, n= 242 | 25 [1 to 209]
  CD20+/27-naive, Yr 2, Wk 24, n= 238 | 21 [2 to 176]
  CD20+/27-naive, Yr 2, Wk 48, n= 224 | 17 [1 to 826]
  CD20+/27-naive, Yr 3, Wk 24, n= 212 | 16 [1 to 243]
  CD20+/27-naive, Yr 3, Wk 48, n= 202 | 14 [1 to 163]
  CD20+/27-naive, Yr 4, Wk 24, n= 196 | 15 [2 to 140]
  CD20+/27-naive, Yr 4, Wk 48, n= 181 | 12 [1 to 152]
  CD20+/27-naive, Yr 5, Wk 24, n= 172 | 12.5 [0 to 127]
  CD20+/27-naive, Yr 5, Wk 48, n= 166 | 11 [2 to 176]
  CD20+/27-naive, Yr 6, Wk 24, n= 159 | 12 [0 to 67]
  CD20+/27-naive, Yr 6, Wk 48, n= 114 | 13 [1 to 68]
  CD20+/27-naive, Yr 7, Wk 24, n= 111 | 13 [1 to 69]
  CD20+/27-naive, Yr 7, Wk 48, n= 87 | 12 [2 to 59]
  CD20+/27-naive, Yr 8, Wk 24, n= 54 | 11.5 [2 to 62]
  CD20+/27-naive, Yr 8, Wk 48, n= 28 | 12 [2 to 54]
  CD20+/27-naive, Yr 9, Wk 24, n= 2 | 5.5 [4 to 7]
  CD20+/27-naive, Exit, n= 207 | 13 [1 to 313]
  CD20+/69+activated, Baseline, n= 257 | 190 [11 to 2492]
  CD20+/69+activated, Yr 1, Wk 24, n= 247 | 131 [7 to 1503]
  CD20+/69+activated, Yr 1, Wk 48, n= 244 | 82 [1 to 561]
  CD20+/69+activated, Yr 2, Wk 24, n= 244 | 74 [0 to 916]
  CD20+/69+activated, Yr 2, Wk 48, n= 233 | 56 [0 to 472]
  CD20+/69+activated, Yr 3, Wk 24, n= 218 | 31 [0 to 242]
  CD20+/69+activated, Yr 3, Wk 48, n= 211 | 22 [0 to 233]
  CD20+/69+activated, Yr 4, Wk 24, n= 210 | 13 [0 to 687]
  CD20+/69+activated, Yr 4, Wk 48, n= 193 | 8 [0 to 288]
  CD20+/69+activated, Yr 5, Wk 24, n= 188 | 6 [0 to 147]
  CD20+/69+activated, Yr 5, Wk 48, n= 181 | 4 [0 to 61]
  CD20+/69+activated, Yr 6, Wk 24, n= 174 | 4 [0 to 40]
  CD20+/69+activated, Yr 6, Wk 48, n= 133 | 3 [0 to 56]
  CD20+/69+activated, Yr 7, Wk 24, n= 122 | 3 [0 to 43]
  CD20+/69+activated, Yr 7, Wk 48, n= 97 | 2 [0 to 29]
  CD20+/69+activated, Yr 8, Wk 24, n= 60 | 1.5 [0 to 21]
  CD20+/69+activated, Yr 8, Wk 48, n= 29 | 1 [0 to 10]
  CD20+/69+activated, Yr 9, Wk 24, n= 2 | 0.5 [0 to 1]
  CD20+/69+activated, Exit, n= 233 | 2 [0 to 457]
  CD20-/138+plasma cells, Baseline, n= 261 | 41 [1 to 870]
  CD20-/138+plasma cells, Yr 1, Wk 24, n= 251 | 31 [0 to 393]
  CD20-/138+plasma cells, Yr 1, Wk 48, n= 247 | 24 [0 to 255]
  CD20-/138+plasma cells, Yr 2, Wk 24, n= 246 | 23 [0 to 446]
  CD20-/138+plasma cells, Yr 2, Wk 48, n= 233 | 20 [0 to 1513]
  CD20-/138+plasma cells, Yr 3, Wk 24, n= 218 | 19 [0 to 312]
  CD20-/138+plasma cells, Yr 3, Wk 48, n= 212 | 16 [0 to 225]
  CD20-/138+plasma cells, Yr 4, Wk 24, n= 211 | 14 [0 to 337]
  CD20-/138+plasma cells, Yr 4, Wk 48, n= 194 | 7.5 [0 to 214]
  CD20-/138+plasma cells, Yr 5, Wk 24, n= 189 | 6 [0 to 135]
  CD20-/138+plasma cells, Yr 5, Wk 48, n= 181 | 6 [0 to 75]
  CD20-/138+plasma cells, Yr 6, Wk 24, n= 174 | 4 [0 to 50]
  CD20-/138+plasma cells, Yr 6, Wk 48, n= 133 | 4 [0 to 64]
  CD20-/138+plasma cells, Yr 7, Wk 24, n= 122 | 4.5 [0 to 84]
  CD20-/138+plasma cells, Yr 7, Wk 48, n= 97 | 4 [0 to 47]
  CD20-/138+plasma cells, Yr 8, Wk 24, n= 60 | 3 [0 to 75]
  CD20-/138+plasma cells, Yr 8, Wk 48, n= 29 | 2 [0 to 28]
  CD20-/138+plasma cells, Yr 9, Wk 24, n= 2 | 8 [2 to 14]
  CD20-/138+plasma cells, Exit, n= 232 | 5 [0 to 221]
  Total CD19+ B-cells (CD19+), Baseline, n= 265 | 114 [4 to 815]
  Total CD19+ B-cells (CD19+), Yr 1, Wk 24, n= 253 | 69 [4 to 437]
  Total CD19+ B-cells (CD19+), Yr 1, Wk 48, n= 254 | 49 [4 to 411]
  Total CD19+ B-cells (CD19+), Yr 2, Wk 24, n= 247 | 37 [4 to 281]
  Total CD19+ B-cells (CD19+), Yr 2, Wk 48, n= 234 | 34 [4 to 1559]
  Total CD19+ B-cells (CD19+), Yr 3, Wk 24, n= 220 | 30 [4 to 296]
  Total CD19+ B-cells (CD19+), Yr 3, Wk 48, n= 212 | 26 [4 to 510]
  Total CD19+ B-cells (CD19+), Yr 4, Wk 24, n= 211 | 25 [4 to 359]
  Total CD19+ B-cells (CD19+), Yr 4, Wk 48, n= 195 | 22 [4 to 245]
  Total CD19+ B-cells (CD19+), Yr 5, Wk 24, n= 190 | 19 [4 to 144]
  Total CD19+ B-cells (CD19+), Yr 5, Wk 48, n= 182 | 18 [4 to 301]
  Total CD19+ B-cells (CD19+), Yr 6, Wk 24, n= 175 | 19 [4 to 117]
  Total CD19+ B-cells (CD19+), Yr 6, Wk 48, n= 132 | 17.5 [4 to 114]
  Total CD19+ B-cells (CD19+), Yr 7, Wk 24, n= 122 | 18.5 [4 to 160]
  Total CD19+ B-cells (CD19+), Yr 7, Wk 48, n= 97 | 19 [4 to 121]
  Total CD19+ B-cells (CD19+), Yr 8, Wk 24, n= 60 | 16.5 [4 to 92]
  Total CD19+ B-cells (CD19+), Yr 8, Wk 48, n= 29 | 15 [4 to 58]
  Total CD19+ B-cells (CD19+), Yr 9, Wk 24, n= 2 | 7.5 [7 to 8]
  Total CD19+ B-cells (CD19+), Exit, n= 234 | 20 [4 to 368]

28. Secondary Outcome: Median Percent Change From Baseline in B Cell Levels at Indicated Time Points.
Description: B-cell levels were assessed at Baseline (BL) (Day 0), Week (Wk) 24 and 48 in first year, at Week 24 and 48 in subsequent years up to 432 weeks and at exit visit. Median percent change from Baseline in absolute B cell subsets (CD20+), CD19+/27BRIGHT/38BRIGHT SLE subset, CD19+20-27hi+ short-lived plasma cells (SLPC), CD20+/138+ plasmacytoid, CD20+/27+ memory, CD20+/27- naïve, CD20+/69+activated, CD20-/138+ plasma cells, Total CD19+ B-cells (CD19+) levels are summarized. The Baseline is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Percent change from Baseline is calculated as: 100 x ([Post-Dose Visit Value - Baseline] / Baseline). Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Week 432
Population: MITT Population
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Percentage change
  CD20+, Yr 1, Wk 24, n= 245 | -31.82 [-91.9 to 394.1]
  CD20+, Yr 1, Wk 48, n= 237 | -51.61 [-94.7 to 216.7]
  CD20+, Yr 2, Wk 24, n= 233 | -61.76 [-95.4 to 250]
  CD20+, Yr 2, Wk 48, n= 218 | -66.21 [-96.3 to 1616.9]
  CD20+, Yr 3, Wk 24, n= 206 | -69.68 [-96.2 to 250]
  CD20+, Yr 3, Wk 48, n= 196 | -72.77 [-97.3 to 270.6]
  CD20+, Yr 4, Wk 24, n= 191 | -75.16 [-96.8 to 82.4]
  CD20+, Yr 4, Wk 48, n= 175 | -78.33 [-97.6 to 561.1]
  CD20+, Yr 5, Wk 24, n= 166 | -80.26 [-97.6 to 156.3]
  CD20+, Yr 5, Wk 48, n= 161 | -81.06 [-98.1 to 93.8]
  CD20+, Yr 6, Wk 24, n= 154 | -81.87 [-98.1 to 2381.3]
  CD20+, Yr 6, Wk 48, n= 109 | -82.94 [-96.7 to 102.9]
  CD20+, Yr 7, Wk 24, n= 107 | -83.22 [-97.6 to 188.9]
  CD20+, Yr 7, Wk 48, n= 82 | -80.96 [-97.3 to 172.2]
  CD20+, Yr 8, Wk 24, n= 52 | -78.94 [-96.9 to 244.4]
  CD20+, Yr 8, Wk 48, n= 27 | -85.29 [-95.5 to 105.9]
  CD20+, Yr 9, Wk 24, n= 2 | -63.65 [-84.4 to -42.9]
  CD20+, Exit, n= 203 | -80.6 [-98.2 to 225]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 1, Wk 24, n= 243 | -16.13 [-100 to 4500]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 1, Wk 48, n= 240 | -38.74 [-100 to 4800]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 2, Wk 24, n= 239 | -25 [-100 to 2200]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 2, Wk 48, n= 225 | -26.23 [-100 to 33100]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 3, Wk 24, n= 210 | -33.97 [-100 to 6800]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 3, Wk 48, n= 204 | -37.98 [-100 to 4900]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 4, Wk 24, n= 204 | -19.52 [-100 to 2787.5]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 4, Wk 48, n= 187 | -16.67 [-100 to 5500]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 5, Wk 24, n= 182 | -33.33 [-100 to 4900]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 5, Wk 48, n= 174 | -37.46 [-100 to 10000]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 6, Wk 24, n= 167 | -44.44 [-100 to 11100]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 6, Wk 48, n= 126 | -50 [-100 to 24700]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 7, Wk 24, n= 117 | -50 [-100 to 29300]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 7, Wk 48, n= 92 | -70.76 [-100 to 2100]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 8, Wk 24, n= 57 | -71.43 [-100 to 1787.5]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 8, Wk 48, n= 28 | -85 [-100 to 100]
  CD19+/27BRIGHT/38BRIGHT SLE, Yr 9, Wk 24, n= 2 | 210.98 [-78 to 500]
  CD19+/27BRIGHT/38BRIGHT SLE, Exit, n= 226 | -50 [-100 to 6100]
  CD19+20-27hi+ SLPC, Yr 1, Wk 24, n= 238 | -32.29 [-100 to 4330]
  CD19+20-27hi+ SLPC, Yr 1, Wk 48, n= 235 | -40 [-100 to 1400]
  CD19+20-27hi+ SLPC, Yr 2, Wk 24, n= 234 | -27.05 [-100 to 2000]
  CD19+20-27hi+ SLPC, Yr 2, Wk 48, n= 221 | -30 [-100 to 4385.7]
  CD19+20-27hi+ SLPC, Yr 3, Wk 24, n= 207 | -37.5 [-100 to 1300]
  CD19+20-27hi+ SLPC, Yr 3, Wk 48, n= 199 | -40.54 [-100 to 6600]
  CD19+20-27hi+ SLPC, Yr 4, Wk 24, n= 199 | -29.41 [-100 to 1900]
  CD19+20-27hi+ SLPC, Yr 4, Wk 48, n= 184 | -29.29 [-100 to 1250]
  CD19+20-27hi+ SLPC, Yr 5, Wk 24, n= 178 | -44.6 [-100 to 1400]
  CD19+20-27hi+ SLPC, Yr 5, Wk 48, n= 171 | -45.65 [-100 to 1328.6]
  CD19+20-27hi+ SLPC, Yr 6, Wk 24, n= 165 | -62.5 [-100 to 3400]
  CD19+20-27hi+ SLPC, Yr 6, Wk 48, n= 123 | -62.5 [-100 to 3400]
  CD19+20-27hi+ SLPC, Yr 7, Wk 24, n= 114 | -47.5 [-100 to 4128.6]
  CD19+20-27hi+ SLPC, Yr 7, Wk 48, n= 89 | -58.33 [-100 to 2900]
  CD19+20-27hi+ SLPC, Yr 8, Wk 24, n= 55 | -62.07 [-100 to 1884.2]
  CD19+20-27hi+ SLPC, Yr 8, Wk 48, n= 27 | -84.62 [-100 to 10.5]
  CD19+20-27hi+ SLPC, Yr 9, Wk 24, n= 1 | -79.4 [-79.4 to -79.4]
  CD19+20-27hi+ SLPC, Exit, n= 224 | -51.42 [-100 to 2000]
  CD20+/138+ plasmacytoid, Yr 1, Wk 24, n= 243 | -32.49 [-97.4 to 6352]
  CD20+/138+ plasmacytoid, Yr 1, Wk 48, n= 240 | -61.11 [-99 to 923.4]
  CD20+/138+ plasmacytoid, Yr 2, Wk 24, n= 239 | -66 [-100 to 2233.3]
  CD20+/138+ plasmacytoid, Yr 2, Wk 48, n= 225 | -70.64 [-99.2 to 422.2]
  CD20+/138+ plasmacytoid, Yr 3, Wk 24, n= 211 | -78.57 [-100 to 644.4]
  CD20+/138+ plasmacytoid, Yr 3, Wk 48, n= 204 | -88.89 [-100 to 863.6]
  CD20+/138+ plasmacytoid, Yr 4, Wk 24, n= 204 | -93.14 [-100 to 156]
  CD20+/138+ plasmacytoid, Yr 4, Wk 48, n= 186 | -94.17 [-100 to 35]
  CD20+/138+ plasmacytoid, Yr 5, Wk 24, n= 181 | -96.25 [-100 to 33.3]
  CD20+/138+ plasmacytoid, Yr 5, Wk 48, n= 174 | -96.75 [-100 to -21.2]
  CD20+/138+ plasmacytoid, Yr 6, Wk 24, n= 167 | -96.53 [-100 to -9.1]
  CD20+/138+ plasmacytoid, Yr 6, Wk 48, n= 126 | -97.96 [-100 to -36.4]
  CD20+/138+ plasmacytoid, Yr 7, Wk 24, n= 117 | -98 [-100 to -33.3]
  CD20+/138+ plasmacytoid, Yr 7, Wk 48, n= 91 | -98.46 [-100 to -40]
  CD20+/138+ plasmacytoid, Yr 8, Wk 24, n= 57 | -98.64 [-100 to -70]
  CD20+/138+ plasmacytoid, Yr 8, Wk 48, n= 28 | -98.68 [-100 to -92.9]
  CD20+/138+ plasmacytoid, Yr 9, Wk 24, n= 2 | -96.15 [-100 to -92.3]
  CD20+/138+ plasmacytoid, Exit, n= 225 | -96.83 [-100 to 610.7]
  CD20+/27+Memory, Yr 1, Wk 24, n= 244 | 87.65 [-97.1 to 1420]
  CD20+/27+Memory, Yr 1, Wk 48, n= 237 | 42.86 [-100 to 800]
  CD20+/27+Memory, Yr 2, Wk 24, n= 233 | 11.11 [-88.9 to 700]
  CD20+/27+Memory, Yr 2, Wk 48, n= 217 | -7.69 [-84.6 to 5616.7]
  CD20+/27+Memory, Yr 3, Wk 24, n= 205 | -23.26 [-100 to 900]
  CD20+/27+Memory, Yr 3, Wk 48, n= 196 | -35.29 [-97.1 to 3000]
  CD20+/27+Memory, Yr 4, Wk 24, n= 191 | -40 [-92.6 to 1400]
  CD20+/27+Memory, Yr 4, Wk 48, n= 175 | -50 [-92.3 to 3166.7]
  CD20+/27+Memory, Yr 5, Wk 24, n= 166 | -50 [-97.7 to 500]
  CD20+/27+Memory, Yr 5, Wk 48, n= 160 | -58.87 [-96 to 800]
  CD20+/27+Memory, Yr 6, Wk 24, n= 153 | -57.89 [-96.2 to 533.3]
  CD20+/27+Memory, Yr 6, Wk 48, n= 108 | -63.4 [-92.9 to 400]
  CD20+/27+Memory, Yr 7, Wk 24, n= 106 | -67.18 [-96.2 to 500]
  CD20+/27+Memory, Yr 7, Wk 48, n= 81 | -71.43 [-92.3 to 400]
  CD20+/27+Memory, Yr 8, Wk 24, n= 52 | -67.03 [-96 to 200]
  CD20+/27+Memory, Yr 8, Wk 48, n= 27 | -64.71 [-88.8 to 600]
  CD20+/27+Memory, Yr 9, Wk 24, n= 2 | -75.96 [-76.9 to -75]
  CD20+/27+Memory, Exit, n= 202 | -61.41 [-100 to 1000]
  CD20+/27-naive, Yr 1, Wk 24, n= 245 | -55.56 [-95.1 to 337.5]
  CD20+/27-naive, Yr 1, Wk 48, n= 237 | -69.7 [-96.7 to 200]
  CD20+/27-naive, Yr 2, Wk 24, n= 233 | -77.27 [-97.6 to 150]
  CD20+/27-naive, Yr 2, Wk 48, n= 218 | -79.5 [-98.6 to 959]
  CD20+/27-naive, Yr 3, Wk 24, n= 206 | -80.11 [-98.5 to 100]
  CD20+/27-naive, Yr 3, Wk 48, n= 196 | -84.41 [-98.5 to 500]
  CD20+/27-naive, Yr 4, Wk 24, n= 191 | -81.93 [-98.8 to 100]
  CD20+/27-naive, Yr 4, Wk 48, n= 175 | -84.21 [-98.8 to 100]
  CD20+/27-naive, Yr 5, Wk 24, n= 166 | -86.09 [-100 to 66.7]
  CD20+/27-naive, Yr 5, Wk 48, n= 161 | -87.5 [-99.2 to 57.7]
  CD20+/27-naive, Yr 6, Wk 24, n= 154 | -86.88 [-100 to 233.3]
  CD20+/27-naive, Yr 6, Wk 48, n= 109 | -86.93 [-97.7 to 100]
  CD20+/27-naive, Yr 7, Wk 24, n= 107 | -87.39 [-98.4 to 300]
  CD20+/27-naive, Yr 7, Wk 48, n= 82 | -84.78 [-98 to 300]
  CD20+/27-naive, Yr 8, Wk 24, n= 52 | -83.7 [-97.9 to 510]
  CD20+/27-naive, Yr 8, Wk 48, n= 27 | -88.15 [-96.5 to 86.7]
  CD20+/27-naive, Yr 9, Wk 24, n= 2 | -61.93 [-87.5 to -36.4]
  CD20+/27-naive, Exit, n= 203 | -86.42 [-99 to 433.3]
  CD20+/69+activated, Yr 1, Wk 24, n= 240 | -33.35 [-98.5 to 3000]
  CD20+/69+activated, Yr 1, Wk 48, n= 238 | -56.33 [-99.7 to 1331.6]
  CD20+/69+activated, Yr 2, Wk 24, n= 236 | -65.21 [-100 to 580]
  CD20+/69+activated, Yr 2, Wk 48, n= 223 | -72.31 [-100 to 502.9]
  CD20+/69+activated, Yr 3, Wk 24, n= 208 | -83.71 [-100 to 306.9]
  CD20+/69+activated, Yr 3, Wk 48, n= 202 | -89.28 [-100 to 325.7]
  CD20+/69+activated, Yr 4, Wk 24, n= 201 | -93.14 [-100 to 89.3]
  CD20+/69+activated, Yr 4, Wk 48, n= 185 | -94.85 [-100 to 263.6]
  CD20+/69+activated, Yr 5, Wk 24, n= 180 | -96.99 [-100 to 13.4]
  CD20+/69+activated, Yr 5, Wk 48, n= 172 | -98.04 [-100 to 14.3]
  CD20+/69+activated, Yr 6, Wk 24, n= 165 | -98.04 [-100 to -16.7]
  CD20+/69+activated, Yr 6, Wk 48, n= 125 | -98.76 [-100 to 20]
  CD20+/69+activated, Yr 7, Wk 24, n= 116 | -98.85 [-100 to -24.1]
  CD20+/69+activated, Yr 7, Wk 48, n=89 | -99.22 [-100 to -76]
  CD20+/69+activated, Yr 8, Wk 24, n= 56 | -99.33 [-100 to -83.7]
  CD20+/69+activated, Yr 8, Wk 48, n= 28 | -99.71 [-100 to -95.8]
  CD20+/69+activated, Yr 9, Wk 24, n= 2 | -97.92 [-100 to -95.8]
  CD20+/69+activated, Exit, n= 226 | -98.99 [-100 to 453.1]
  CD20-/138+plasma cells, Yr 1, Wk 24, n= 244 | -37.2 [-100 to 3400]
  CD20-/138+plasma cells, Yr 1, Wk 48, n= 241 | -50 [-100 to 4700]
  CD20-/138+plasma cells, Yr 2, Wk 24, n= 240 | -47.83 [-100 to 1200]
  CD20-/138+plasma cells, Yr 2, Wk 48, n= 226 | -53.92 [-100 to 5500]
  CD20-/138+plasma cells, Yr 3, Wk 24, n= 212 | -64.82 [-100 to 1000]
  CD20-/138+plasma cells, Yr 3, Wk 48, n= 205 | -71.43 [-100 to 2566.7]
  CD20-/138+plasma cells, Yr 4, Wk 24, n= 205 | -73.76 [-100 to 910]
  CD20-/138+plasma cells, Yr 4, Wk 48, n= 187 | -81.58 [-100 to 586.4]
  CD20-/138+plasma cells, Yr 5, Wk 24, n= 182 | -86.46 [-100 to 133.3]
  CD20-/138+plasma cells, Yr 5, Wk 48, n= 175 | -88.89 [-100 to 300]
  CD20-/138+plasma cells, Yr 6, Wk 24, n= 168 | -91.3 [-100 to 900]
  CD20-/138+plasma cells, Yr 6, Wk 48, n= 127 | -90.91 [-100 to 2100]
  CD20-/138+plasma cells, Yr 7, Wk 24, n= 118 | -92.31 [-100 to 1700]
  CD20-/138+plasma cells, Yr 7, Wk 48, n= 92 | -93.83 [-100 to 200]
  CD20-/138+plasma cells, Yr 8, Wk 24, n= 57 | -93.39 [-100 to -11.1]
  CD20-/138+plasma cells, Yr 8, Wk 48, n= 28 | -97.56 [-100 to -75]
  CD20-/138+plasma cells, Yr 9, Wk 24, n= 2 | -80.78 [-90.1 to -71.4]
  CD20-/138+plasma cells, Exit, n= 226 | -88.58 [-100 to 1600]
  Total CD19+ B-cells (CD19+), Yr 1, Wk 24, n= 250 | -32.56 [-91.7 to 400]
  Total CD19+ B-cells (CD19+), Yr 1, Wk 48, n= 251 | -51.61 [-94.6 to 214.3]
  Total CD19+ B-cells (CD19+), Yr 2, Wk 24, n= 244 | -61.71 [-95.5 to 244.4]
  Total CD19+ B-cells (CD19+), Yr 2, Wk 48, n= 231 | -66.67 [-96 to 1576.3]
  Total CD19+ B-cells (CD19+), Yr 3, Wk 24, n= 217 | -70.21 [-96.3 to 153.3]
  Total CD19+ B-cells (CD19+), Yr 3, Wk 48, n= 209 | -74.24 [-97.3 to 276.5]
  Total CD19+ B-cells (CD19+), Yr 4, Wk 24, n= 209 | -75.61 [-97.8 to 82.4]
  Total CD19+ B-cells (CD19+), Yr 4, Wk 48, n= 192 | -78.54 [-97.8 to 528.2]
  Total CD19+ B-cells (CD19+), Yr 5, Wk 24, n= 187 | -80.56 [-97.8 to 141.2]
  Total CD19+ B-cells (CD19+), Yr 5, Wk 48, n= 179 | -81.14 [-98.1 to 100]
  Total CD19+ B-cells (CD19+), Yr 6, Wk 24, n= 172 | -81.85 [-98.1 to 75]
  Total CD19+ B-cells (CD19+), Yr 6, Wk 48, n= 130 | -82.34 [-98.5 to 79.5]
  Total CD19+ B-cells (CD19+), Yr 7, Wk 24, n= 120 | -82.73 [-97.6 to 125]
  Total CD19+ B-cells (CD19+), Yr 7, Wk 48, n= 95 | -80.95 [-97.8 to 172.2]
  Total CD19+ B-cells (CD19+), Yr 8, Wk 24, n= 59 | -79.87 [-96.9 to 250]
  Total CD19+ B-cells (CD19+), Yr 8, Wk 48, n= 28 | -84.79 [-95.6 to 94.4]
  Total CD19+ B-cells (CD19+), Yr 9, Wk 24, n= 2 | -66.04 [-85.4 to -46.7]
  Total CD19+ B-cells (CD19+), Exit, n= 232 | -80.81 [-98.2 to 178.6]

29. Secondary Outcome: Percentage of Participants With Worsening in SLICC/ACR Damage Index at Indicated Time Points
Description: Systemic Lupus International Collaborative Clinics/American College of Rheumatology (SLICC/ACR) Damage Index is a tool used to assess non-reversible organ damage in SLE patients. Damage Index is used to assess 12 systems by 41 items. Score is given as 1 or sometimes 2, if occur more than once, so that that the maximum possible score is 47. Higher damage index scores early in disease are associated with a poor prognosis and with increased mortality. Damage index was assessed at BL (Day 0), Week 48 in first year, at Week 48 in subsequent years up to 8 years. Percentage of participants with worsening in damage index (change >0) are summarized. The BL is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Only those participants available at the specified time points were analyzed ( n=X).
Time Frame: Up to Week 384
Population: MITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Percentage of Participants
  Year 1, Week 48, n=263 | 5.7
  Year 2, Week 48, n=256 | 12.1
  Year 3, Week 48, n=239 | 18
  Year 4, Week 48, n=212 | 20.8
  Year 5, Week 48, n=195 | 22.6
  Year 6, Week 48, n=187 | 25.1
  Year 7, Week 48, n=126 | 30.2
  Year 8, Week 48, n=65 | 29.2

30. Secondary Outcome: Change From Baseline in SF-36 Healthy Survey Overall Component Scores at Indicated Time Point
Description: The SF-36v2 is a participant-reported short form survey to measure functional health and well-being. There are 36 items grouped into eight health domains: Vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. SF-36v2 gives a score (0-100) for each of these domains as well as summary score for the physical component score (PCS) and mental component score (MCS) based on the responses by participants. The lower the score the more disability and the higher the score the less disability. The BL is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from BL was calculated as the individual post-BL value minus the BL value. Only those participants available at the specified time points were analyzed ( n=X).
Time Frame: Up to Week 384
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Score on a scale
  MCS, Year 1, Week 48, n= 259 | 2.47 (10.113)
  MCS, Year 2, Week 48, n= 255 | 2.99 (10.428)
  MCS, Year 3, Week 48, n= 236 | 2.54 (10.399)
  MCS, Year 4, Week 48, n= 212 | 2.52 (11.099)
  MCS, Year 5, Week 48, n= 193 | 2.22 (11.22)
  MCS, Year 6, Week 48, n= 185 | 2.71 (11.274)
  MCS, Year 7, Week 48, n= 126 | 3.19 (11.269)
  MCS, Year 8, Week 48, n= 65 | 3.91 (11.066)
  PCS, Year 1, Week 48, n= 259 | 3.41 (8.603)
  PCS, Year 2, Week 48, n= 255 | 4.64 (8.3)
  PCS, Year 3, Week 48, n= 236 | 5.93 (8.51)
  PCS, Year 4, Week 48, n= 212 | 5.01 (8.752)
  PCS, Year 5, Week 48, n= 193 | 6.12 (9.314)
  PCS, Year 6, Week 48, n= 185 | 4.79 (9.406)
  PCS, Year 7, Week 48, n= 126 | 7.7 (9.887)
  PCS, Year 8, Week 48, n= 65 | 6.73 (10.107)

31. Secondary Outcome: Change From Baseline in SF-36 Healthy Survey Overall Component Scores at Indicated Timepoints
Description: The SF-36v2 is a participant-reported survey to measure functional health and well-being. There are 36 items grouped into eight health domains: Vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. SF-36v2 gives a score (0-100) for each of these domains as well as summary score for the physical component score (PCS) and mental component score (MCS) based on the responses by participants. The lower the score the more disability and the higher the score the less disability. The BL is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from BL was calculated as the individual post-BL value minus the BL value. Only those participants available at the specified time points were analyzed ( n=X).
Time Frame: Up to Week 384
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Score on a scale
  Bodily pain, Year 1 , Week 48, n= 261 | 9.7 (23.36)
  Bodily pain, Year 2 , Week 48, n= 255 | 9.2 (24.389)
  Bodily pain, Year 3 , Week 48, n= 236 | 10.97 (23.409)
  Bodily pain, Year 4 , Week 48, n= 212 | 8.33 (24.181)
  Bodily pain, Year 5 , Week 48, n= 193 | 10.88 (24.549)
  Bodily pain, Year 6 , Week 48, n= 185 | 8.82 (23.636)
  Bodily pain, Year 7 , Week 48, n= 126 | 14.48 (24.969)
  Bodily pain, Year 8 , Week 48, n= 65 | 11.94 (22.93)
  General health, Year 1 , Week 48, n= 260 | 5.66 (14.693)
  General health, Year 2 , Week 48, n= 255 | 6.14 (15.156)
  General health, Year 3 , Week 48, n= 236 | 8.84 (15.929)
  General health, Year 4 , Week 48, n= 212 | 7.29 (16.069)
  General health, Year 5 , Week 48, n= 193 | 9.19 (17.742)
  General health, Year 6 , Week 48, n= 185 | 7.24 (18.187)
  General health, Year 7 , Week 48, n= 126 | 8.71 (18.693)
  General health, Year 8 , Week 48, n= 65 | 8.18 (19.994)
  Mental health, Year 1 , Week 48, n= 260 | 4 (17.71)
  Mental health, Year 2 , Week 48, n= 255 | 3.62 (17.46)
  Mental health, Year 3 , Week 48, n= 236 | 2.34 (17.817)
  Mental health, Year 4 , Week 48, n= 212 | 2.33 (20.172)
  Mental health, Year 5 , Week 48, n= 193 | 1.78 (20.662)
  Mental health, Year 6 , Week 48, n= 185 | 3.6 (19.968)
  Mental health, Year 7 , Week 48, n= 126 | 4.39 (19.811)
  Mental health, Year 8 , Week 48, n= 65 | 6.08 (18.551)
  Physical functioning, Year 1 , Week 48, n= 260 | 6.34 (21.498)
  Physical functioning, Year 2 , Week 48, n= 255 | 6.25 (21.185)
  Physical functioning, Year 3 , Week 48, n= 236 | 7.85 (21.994)
  Physical functioning, Year 4 , Week 48, n= 212 | 6.38 (22.112)
  Physical functioning, Year 5 , Week 48, n= 193 | 7.62 (24.486)
  Physical functioning, Year 6 , Week 48, n= 185 | 6.72 (24.81)
  Physical functioning, Year 7 , Week 48, n= 126 | 11.25 (26.422)
  Physical functioning, Year 8 , Week 48, n= 65 | 11.83 (27.065)
  Role emotional, Year 1 , Week 48, n= 261 | 4.96 (25.714)
  Role emotional, Year 2 , Week 48, n= 254 | 4.74 (27.92)
  Role emotional, Year 3 , Week 48, n= 236 | 3.73 (28.258)
  Role emotional, Year 4 , Week 48, n= 212 | 3.32 (28.237)
  Role emotional, Year 5 , Week 48, n= 193 | 3.61 (28.774)
  Role emotional, Year 6 , Week 48, n= 185 | 3.13 (31.614)
  Role emotional, Year 7 , Week 48, n= 126 | 3.27 (30.385)
  Role emotional, Year 8 , Week 48, n=65 | 7.18 (33.91)
  Role physical, Year 1 , Week 48, n= 260 | 8.91 (26.393)
  Role physical, Year 2 , Week 48, n= 253 | 8 (27.106)
  Role physical, Year 3 , Week 48, n= 236 | 10.05 (26.525)
  Role physical, Year 4 , Week 48, n= 212 | 8.27 (28.998)
  Role physical, Year 5 , Week 48, n= 193 | 10.86 (29.839)
  Role physical, Year 6 , Week 48, n= 185 | 6.91 (30.995)
  Role physical, Year 7 , Week 48, n= 126 | 13.53 (31.347)
  Role physical, Year 8 , Week 48, n= 65 | 11.51 (34.385)
  Social functioning, Year 1 , Week 48, n= 261 | 7.61 (26.901)
  Social functioning, Year 2 , Week 48, n= 255 | 7.21 (27.218)
  Social functioning, Year 3 , Week 48, n= 236 | 9.59 (27.989)
  Social functioning, Year 4 , Week 48, n= 212 | 6.9 (28.598)
  Social functioning, Year 5 , Week 48, n= 193 | 8.16 (30.079)
  Social functioning, Year 6 , Week 48, n= 185 | 6.96 (28.695)
  Social functioning, Year 7 , Week 48, n= 126 | 10.32 (31.784)
  Social functioning, Year 8 , Week 48, n= 65 | 9.81 (32.135)
  Vitality, Year 1 , Week 48, n= 260 | 8.87 (21.449)
  Vitality, Year 2 , Week 48, n= 255 | 7.13 (22.287)
  Vitality, Year 3 , Week 48, n= 236 | 8.17 (20.742)
  Vitality, Year 4 , Week 48, n= 212 | 8.04 (21.742)
  Vitality, Year 5 , Week 48, n= 193 | 8.23 (24.937)
  Vitality, Year 6 , Week 48, n= 185 | 6.93 (23.023)
  Vitality, Year 7 , Week 48, n= 126 | 11.69 (22.709)
  Vitality, Year 8 , Week 48, n= 65 | 6.47 (22.033)

32. Secondary Outcome: Change From Baseline in FACIT-Fatigue Scale Total Score at Indicated Time Point
Description: The FACIT-F scale measures the severity and impact of fatigue on functioning and health related quality of life experienced in the past 7 days. FACIT-Fatigue scale total score was assessed at BL (Day 0), Wk 48 in first year, at Wk 48 in subsequent Yrs up to 8 Yrs.The level of fatigue is measured by 13 questions assessed on a four-point scale (0=not at all fatigued; 1=a little bit fatigued; 2=somewhat fatigued; 3=quite a bit fatigued; 4=very much fatigued; possible total score of 0 to 52). Change from BL in FACIT-Fatigue scale total score are summarized. The BL is defined as the Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from BL was calculated as the individual post-BL value minus the BL value. A negative change from BL represents a worsening condition. Only those participants available at the specified time points were analyzed ( n=X).
Time Frame: Up to Week 384
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Score on a scale
  Year 1, Week 48, n= 260 | 4.91 (10.785)
  Year 2, Week 48, n= 252 | 4.82 (11.414)
  Year 3, Week 48, n= 235 | 4.85 (11.614)
  Year 4, Week 48, n= 210 | 4.14 (11.269)
  Year 5, Week 48, n= 193 | 4.81 (11.962)
  Year 6, Week 48, n= 184 | 3.7 (11.787)
  Year 7, Week 48, n= 126 | 5.74 (11.644)
  Year 8, Week 48, n= 65 | 4.28 (10.949)

33. Secondary Outcome: Percentage of Participants With Improvement in FACIT-Fatigue Scale Score Exceeding the MCID at Indicated Time Points
Description: The FACIT-F scale measures the severity and impact of fatigue on functioning and health related quality of life experienced in the past 7 days. FACIT-Fatigue scale total score was assessed at BL (Day 0), Week 48 in first year, at Week 48 in subsequent years up to 8 years. The level of fatigue is measured by 13 questions assessed on a four-point scale (0=not at all fatigued; 1=a little bit fatigued; 2=somewhat fatigued; 3=quite a bit fatigued; 4=very much fatigued; possible total score of 0 to 52). Percentage of participants with improvement in FACIT-Fatigue scale score exceeding the minimum clinically important difference (MCID) (>=4 points) are summarized. Only those participants available at the specified time points were analyzed ( n=X).
Time Frame: Up to Week 384
Population: MITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 268
Percentage of Participants
  Year 1, Week 48 | 50.4
  Year 2, Week 48 | 45.9
  Year 3, Week 48 | 44.4
  Year 4, Week 48 | 36.2
  Year 5, Week 48 | 40.3
  Year 6, Week 48 | 33.2
  Year 7, Week 48 | 26.1
  Year 8, Week 48 | 13.1

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from Day 1 until follow-up (up to Week 440).
Description: SAEs and non-serious AEs were collected in members of the MITT Population, comprised of all participants who received at least one dose of study medication.
Groups:
- Belimumab 10 mg/kg IV: Belimumab 10 mg/kg IV every 28 days
Arm/Group | Belimumab 10 mg/kg IV
Serious Adverse Events (participants affected / at risk) | 112/268
Other Adverse Events (participants affected / at risk) | 266/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab 10 mg/kg IV (N=268)
Any event (Infections and infestations) | 44
Cellulitis (Infections and infestations) | 7
Pneumonia (Infections and infestations) | 5
Pneumonia bacterial (Infections and infestations) | 5
Gastroenteritis viral (Infections and infestations) | 3
Pneumonia viral (Infections and infestations) | 3
Bacterial pyelonephritis (Infections and infestations) | 2
Bronchitis bacterial (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Cellulitis staphylococcal (Infections and infestations) | 1
Cellulitis streptococcal (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infected dermal cyst (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pelvic abscess (Infections and infestations) | 1
Perinephric abscess (Infections and infestations) | 1
Pharyngitis bacterial (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Staphylococcal skin infection (Infections and infestations) | 1
Streptococcal urinary tract infection (Infections and infestations) | 1
Sweat gland infection (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Any event (Musculoskeletal and connective tissue disorders) | 22
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Any event (General disorders) | 20
Non-cardiac chest pain (General disorders) | 12
Pyrexia (General disorders) | 5
Chest pain (General disorders) | 2
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Any event (Gastrointestinal disorders) | 19
Abdominal pain (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Abdominal adhesions (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Oesophageal spasm (Gastrointestinal disorders) | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Any event (Injury, poisoning and procedural complications) | 15
Procedural haemorrhage (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 2
Post procedural complication (Injury, poisoning and procedural complications) | 2
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Any event (Nervous system disorders) | 15
Syncope (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Amnesia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Any event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oestrogen receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Any event (Respiratory, thoracic and mediastinal disorders) | 11
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Any event (Vascular disorders) | 10
Hypertension (Vascular disorders) | 3
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Lupus vasculitis (Vascular disorders) | 1
Malignant hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1
Subgaleal haematoma (Vascular disorders) | 1
Any event (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Any event (Cardiac disorders) | 7
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Hypertensive heart disease (Cardiac disorders) | 1
Mitral valve disease (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Any event (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 1
Dysthymic disorder (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Any event (Renal and urinary disorders) | 7
Lupus nephritis (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 2
Calculus ureteric (Renal and urinary disorders) | 1
Hypertonic bladder (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Any event (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 2
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Any event (Hepatobiliary disorders) | 5
Cholelithiasis (Hepatobiliary disorders) | 4
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Any event (Reproductive system and breast disorders) | 4
Uterovaginal prolapse (Reproductive system and breast disorders) | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Cystocele (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Any event (Immune system disorders) | 2
Drug hypersensitivity (Immune system disorders) | 2
Any event (Skin and subcutaneous tissue disorders) | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1
Any event (Congenital, familial and genetic disorders) | 1
Spinocerebellar ataxia (Congenital, familial and genetic disorders) | 1
Any event (Endocrine disorders) | 1
Thyroid mass (Endocrine disorders) | 1
Any event (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Any event (Investigations) | 1
Influenza A virus test positive (Investigations) | 1
Influenza B virus test positive (Investigations) | 1
Any event (Pregnancy, puerperium and perinatal conditions) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab 10 mg/kg IV (N=268)
Any event (Infections and infestations) | 243
Upper respiratory tract infection bacterial (Infections and infestations) | 77
Viral upper respiratory tract infection (Infections and infestations) | 76
Urinary tract infection bacterial (Infections and infestations) | 69
Sinusitis (Infections and infestations) | 62
Upper respiratory tract infection (Infections and infestations) | 59
Gastroenteritis viral (Infections and infestations) | 56
Urinary tract infection (Infections and infestations) | 52
Nasopharyngitis (Infections and infestations) | 42
Influenza (Infections and infestations) | 38
Bronchitis bacterial (Infections and infestations) | 36
Vulvovaginal mycotic infection (Infections and infestations) | 36
Bronchitis (Infections and infestations) | 35
Herpes zoster (Infections and infestations) | 24
Cellulitis (Infections and infestations) | 21
Gastroenteritis (Infections and infestations) | 20
Oral herpes (Infections and infestations) | 19
Oral candidiasis (Infections and infestations) | 17
Tooth abscess (Infections and infestations) | 15
Any event (Musculoskeletal and connective tissue disorders) | 217
Arthralgia (Musculoskeletal and connective tissue disorders) | 106
Back pain (Musculoskeletal and connective tissue disorders) | 63
Pain in extremity (Musculoskeletal and connective tissue disorders) | 55
SLE arthritis (Musculoskeletal and connective tissue disorders) | 43
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 41
Bursitis (Musculoskeletal and connective tissue disorders) | 36
Myalgia (Musculoskeletal and connective tissue disorders) | 35
Joint swelling (Musculoskeletal and connective tissue disorders) | 31
Tendonitis (Musculoskeletal and connective tissue disorders) | 27
Muscle spasms (Musculoskeletal and connective tissue disorders) | 26
Neck pain (Musculoskeletal and connective tissue disorders) | 25
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 24
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 22
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 14
Any event (Gastrointestinal disorders) | 191
Nausea (Gastrointestinal disorders) | 86
Diarrhoea (Gastrointestinal disorders) | 58
Vomiting (Gastrointestinal disorders) | 45
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 39
Abdominal pain (Gastrointestinal disorders) | 34
Constipation (Gastrointestinal disorders) | 25
Dental caries (Gastrointestinal disorders) | 21
Mouth ulceration (Gastrointestinal disorders) | 21
Abdominal pain upper (Gastrointestinal disorders) | 20
Dyspepsia (Gastrointestinal disorders) | 18
Any event (Skin and subcutaneous tissue disorders) | 163
Rash (Skin and subcutaneous tissue disorders) | 39
Alopecia (Skin and subcutaneous tissue disorders) | 23
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 22
Pruritus (Skin and subcutaneous tissue disorders) | 20
Dermatitis contact (Skin and subcutaneous tissue disorders) | 16
Eczema (Skin and subcutaneous tissue disorders) | 16
Rash pruritic (Skin and subcutaneous tissue disorders) | 15
Any event (Nervous system disorders) | 162
Headache (Nervous system disorders) | 84
Dizziness (Nervous system disorders) | 29
Migraine (Nervous system disorders) | 25
Hypoaesthesia (Nervous system disorders) | 18
Paraesthesia (Nervous system disorders) | 16
Any event (Injury, poisoning and procedural complications) | 155
Fall (Injury, poisoning and procedural complications) | 44
Ligament sprain (Injury, poisoning and procedural complications) | 27
Contusion (Injury, poisoning and procedural complications) | 25
Procedural pain (Injury, poisoning and procedural complications) | 24
Muscle strain (Injury, poisoning and procedural complications) | 19
Laceration (Injury, poisoning and procedural complications) | 14
Road traffic accident (Injury, poisoning and procedural complications) | 14
Any event (Respiratory, thoracic and mediastinal disorders) | 154
Cough (Respiratory, thoracic and mediastinal disorders) | 51
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 28
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 17
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 16
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 16
Any event (General disorders) | 151
Fatigue (General disorders) | 60
Non-cardiac chest pain (General disorders) | 31
Peripheral swelling (General disorders) | 31
Oedema peripheral (General disorders) | 30
Pyrexia (General disorders) | 30
Pain (General disorders) | 18
Any event (Psychiatric disorders) | 107
Insomnia (Psychiatric disorders) | 57
Anxiety (Psychiatric disorders) | 42
Depression (Psychiatric disorders) | 30
Any event (Metabolism and nutrition disorders) | 89
Vitamin D deficiency (Metabolism and nutrition disorders) | 34
Hypokalaemia (Metabolism and nutrition disorders) | 17
Any event (Investigations) | 86
Weight increased (Investigations) | 25
Any event (Vascular disorders) | 85
Hypertension (Vascular disorders) | 44
Any event (Eye disorders) | 79
Cataract (Eye disorders) | 18
Any event (Cardiac disorders) | 56
Palpitations (Cardiac disorders) | 20
Any event (Immune system disorders) | 53
Seasonal allergy (Immune system disorders) | 29
Drug hypersensitivity (Immune system disorders) | 17
Any event (Ear and labyrinth disorders) | 37
Vertigo (Ear and labyrinth disorders) | 16
Sinusitis bacterial (Infections and infestations) | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.